CLINICAL TRIAL: NCT00655824
Title: An Open-label, International, Multi-center, Phase II, Extension Trial Investigating Long-term Efficacy and Safety of Repeated Treatment Courses of Ofatumumab, a Fully Human Monoclonal Anti-CD20 Antibody, in Adult Patients With Active Rheumatoid Arthritis Who Previously Received Ofatumumab or Placebo
Brief Title: Long-term Efficacy and Safety of Repeated Ofatumumab Treatment Courses in RA Patients Who Previously Received Ofatumumab or Placebo in Trial Hx-CD20-403
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The clinical development of intravenously administered ofatumumab in RA will no longer be pursued, so this study was prematurely terminated by the Sponsor.
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 111752; GEN413 (Other: GENMAB)
Record Dates: First submitted 2008-04-04; First posted 2008-04-10 (Estimated); Results first posted 2012-04-18 (Estimated); Last update posted 2017-12-05 (Actual); Status verified 2017-10

CONDITIONS: Arthritis, Rheumatoid
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ofatumumab (Experimental): 1000 mL dilution of 35mls ofatumumab in sterile, pyrogen free, 0.9% NaCl
  Interventions: Drug: ofatumumab

INTERVENTIONS:
Drug: ofatumumab — 1000 mL dilution of 35mls ofatumumab in sterile, pyrogen free, 0.9% NaCl

SUMMARY:
A 3-year open-label trial for patients who previously participated in Trial Hx-CD20-403 and who fulfill the eligibility criteria for this trial (GEN413) . Th e primary purpose of the trial is to evaluate the long-term effectiveness of repeated courses ( a maximum of 9 treatment courses) of ofatumumab in RA patients who previously received ofatumumab or placebo in Trial Hx-CD20-403.

DETAILED DESCRIPTION:
All patients who fulfill the eligibility criteria for this trial , will initiate at least one treatment course of ofatumumab, and depending of subsequent worsening in disease activity will be eligible to received further treatment through the 156 week treatment period: a maximum of a further 8 treatment courses will be given at individualized time intervals . The interval between each treatment course will be at least 16 weeks with the last treatment course given no later than week 130 after baseline (Visit 2A).

After each treatment course the patients will attend their next trial visit 8 weeks after Infusion 1, followed by trial visits every 4 weeks up to Week 24, and subsequently every 8 weeks until the next treatment course.

After completing the Treatment Period or after withdrawing from the Treatment Period prematurely patients will be followed every 12 weeks (Follow-up Period) until CD19+ cells &/or IgG levels have returned to baseline or normal levels.

ELIGIBILITY:
Inclusion Criteria:

* Previously received ofatumumab or placebo in Trial Hx-CD20-403.
* Patients on methotrexate therapy (7.5 - 25 mg/week, p.o., i.m., and/or s.c.).
* Oral corticosteroids therapy (≤ 10 mg/day prednisolone or equivalent).
* Active disease at the time of screening as defined by:

  * 3 swollen joints (of 28 joints assessed) and ≥ 3 tender joints (of 28 joints assessed), DAS28≥3.2 (based on ESR)

Exclusion Criteria:

* Use of DMARDs other than methotrexate or exposure to other cell depleting therapy, including investigational compounds < 6 months prior to Visit 2 A.
* Patients who have received treatment with any non-marketed drug substance within 4 weeks prior to Visit 1 (screening).
* Breast feeding women or women with a positive pregnancy test at Visit 1 (screening).
* Received anti-cancer therapy, corticosteroids (intra-articular, i.m., or i.v.), or live/attenuated vaccinations, or exposure to cyclophosphamide, nitrogen mustard, chlorambucil or other alkylating agents < 5 years prior to screening.
* Past or current malignancy, except for Cervical carcinoma Stage 1B or less, Non-invasive basal cell and squamous cell skin carcinoma, Malignant melanoma with a complete response of a duration of > 10 years, or other cancer diagnoses with a complete response of a duration of > 5 years.
* Chronic or ongoing active infectious disease requiring systemic treatment.
* Clinically significant cardiac disease, or history of significant cerebrovascular disease.

Significant concurrent, uncontrolled medical conditions, but not limited to, renal, hepatic, hematological, gastrointestinal, endocrine, pulmonary, neurological, cerebral psychiatric disease

* Known or suspected HIV positive, positive serology for hepatitis B (HB), positive test for Hepatitis C, or positive plasma or white cell JC virus (JCV) PCR (either compartment).
* A circulating IgG level <lower limit of normal.
* Known hypersensitivity to components of the investigational medicinal product.
* Patients known or suspected of not being able to comply with a study protocol.
* Women of child bearing potential not will to use adequate contraception during study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2008-01-01; Primary Completion 2011-05-25 (Actual); Study Completion 2013-03-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (10):
- United States (4):
  - GSK Investigational Site, Los Angeles, California
  - GSK Investigational Site, Fort Lauderdale, Florida
  - GSK Investigational Site, New York, New York
  - GSK Investigational Site, Duncansville, Pennsylvania
- Denmark (3):
  - GSK Investigational Site, Copenhagen
  - GSK Investigational Site, Glostrup Municipality
  - GSK Investigational Site, Hellerup
- GSK Investigational Site, Szombathely, Hungary
- GSK Investigational Site, Warsaw, Poland
- GSK Investigational Site, Ipswich, United Kingdom

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants who previously participated in Study OFA112657 (NCT00291928) and who fulfilled the eligibility criteria were offered participation in this study (111752; NCT00655824).
Pre-assignment Details: A participant was considered to have completed the study when the Investigator decided that the participant had completed the treatment phase and recorded this in the Case Report Form. Completion was not based on having completed a set number of treatment courses.
Groups:
- Ofatumumab 700 mg IV Infusion: Ofatumumab was administered in the dose of 700 milligrams (mg) as two intravenous (IV) infusions separated by 2 weeks for the first treatment course. The remaining treatment courses were given at individualized time intervals when a clinical response had been achieved following the previous treatment course and a subsequent worsening in disease activity had been observed. For the remaining treatment courses, the interval between the treatment courses was at least 16 weeks from the first infusion in the previous treatment course irrespective of progression in disease activity. After each treatment course, the participants attended their next trial visit 8 weeks after the first infusion of that course, followed by trial visits every 4 weeks up to Week 24, and subsequent visits every 8 weeks until the next treatment course. A maximum of 9 treatment courses were allowed.
Period: Overall Study
Arm/Group | Ofatumumab 700 mg IV Infusion
Started | 92
Completed | 8
Not Completed | 84
Not completed — Adverse Event | 3
Not completed — Early Termination of Study by Sponsor | 74
Not completed — Protocol Violation | 1
Not completed — Withdrawal by Subject | 4
Not completed — Deterioration of Trial Disease | 2

BASELINE CHARACTERISTICS:
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
Age, Continuous [Mean (Standard Deviation); unit: Years] | 52.9 (10.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 84
  Male | 8
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 92

OUTCOME MEASURES:

1. Primary Outcome: Time to Treatment Withdrawal
Description: Time to treatment withdrawal was defined as the time from the first infusion of ofatumumab until the date of treatment withdrawal. The sponsor discontinued the intravenous route of administration development program for rheumatoid arthritis (RA), and this study was terminated early; hence, this primary endpoint was not evaluated.
Time Frame: From Baseline up to 144 weeks
Population: Full Analysis Set (FAS) Population: all participants who were exposed to study drug irrespective of their compliance to the planned course of treatment.
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 0

2. Secondary Outcome: Minimum Change From Baseline in Disease Activity Score Based on 28 Joints (DAS28) Over the Course of Weeks (Wk) 1 to 24 in Each Treatment Course (TC), Assessed by Erythrocyte Sedimentation Rate (ESR; Rate at Which Red Blood Cells Sediment in 1 Hour)
Description: DAS28(ESR) is a numeric outcome that measures RA activity based on the ESR (a non-specific general indicator of inflammation), tender joint count (JC), swollen JC, and participant's global assessment of disease activity on a 100 millimeter Visual Analog Scale. DAS28 values range from 0 (no activity) and upwards; increasing values indicate increasing activity (there is no upper limit on the scale). Change from baseline (CFB) was calculated at all visits; however, minimum CFB was calculated as the minimum CFB obtained over the course of weeks 1-24 of each treatment cycle.
Time Frame: Baseline (last visit prior to dosing in each TC) and last visit of each TC (8 wk post infusion, then every 4 wk until Wk 24; up to 144 weeks). TCs were individualized based on clinical status and may not correlate to trial visits or study weeks.
Population: FAS Population. One participant withdrew during the first infusion due to adverse events (AEs) of rash and pruritus. Only participants available at the indicated time point were assessed. Minimum change from baseline is defined as the smallest change at any visit over the course of Weeks 1 to 24 of each treatment cycle.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 91
scores on a scale
  Treatment Course 1, n=91 | -1.92 (0.918)
  Treatment Course 2, n=71 | -1.58 (0.824)
  Treatment Course 3, n=53 | -1.52 (0.849)
  Treatment Course 4, n=20 | -1.65 (1.110)
  Treatment Course 5, n=8 | -2.16 (1.114)
  Treatment Course 6, n=4 | -0.87 (0.771)
  Treatment Course 7, n=2 | -2.10 (2.146)

3. Secondary Outcome: Minimum Change From Baseline in DAS28 Over the Course of Weeks 1 to 24 in Each Treatment Course, Based on C-reactive Protein (CRP)
Description: DAS28(CRP) is a numeric outcome that measures RA activity based on the CRP (used to monitor acute inflammatory phases of RA), tender JC, swollen JC, and participant's global assessment of disease activity on a 100 millimeter Visual Analog Scale. DAS28 values range from 0 (no activity) and upwards; increasing values indicate increasing activity (there is no upper limit on the scale). Change from baseline (CFB) was calculated at all visits; however, minimum CFB was calculated as the minimum CFB obtained over the course of weeks 1-24 of each treatment cycle.
Time Frame: as for outcome 2
Population: FAS Population. One participant withdrew during the first infusion due to AEs of rash and pruritis. Only participants available at the indicated time point were assessed.
Measure: Mean (Standard Deviation); unit: scores on a scale
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 91
scores on a scale
  Treatment Course 1, n=91 | -1.79 (0.906)
  Treatment Course 2, n=71 | -1.32 (0.771)
  Treatment Course 3, n=53 | -1.27 (0.793)
  Treatment Course 4, n=20 | -1.55 (0.970)
  Treatment Course 5, n=8 | -1.88 (1.181)
  Treatment Course 6, n=4 | -0.88 (0.572)
  Treatment Course 7, n=2 | -2.14 (1.893)

4. Secondary Outcome: Time to Re-treatment in Each Treatment Course
Description: Time to re-treatment in each treatment course (TC) is defined as the time from the first infusion of ofatumumab until the date of the first infusion of the first re-treatment course. The data presented reflect the time to re-treatment, which is defined as the time in days between the first infusion of each TC and the first infusion of the following TC. For TC 1, time to re-treatment is defined as the time between the first infusion in TC 1 and the first infusion in TC 2; similarly, for TC 2 it is the time between the first infusion of TC 2 and the first infusion of TC 3. The study was terminated by the sponsor after Treatment Course 7; therefore, there are no re-treatment data available for Treatment Course 7.
Time Frame: Week 16 to Week 104 of each treatment course (up to 125 weeks). TCs were individualized based on clinical status and may not correlate to trial visits or study weeks.
Population: FAS Population. Only participants available at the indicated time point were assessed.
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 73
days
  Treatment Course 1, n=73 | 291.01 (127.367)
  Treatment Course 2, n=53: number analyzed (Participants) | 53
  Treatment Course 2, n=53 | 328.83 (122.427)
  Treatment Course 3, n=20: number analyzed (Participants) | 20
  Treatment Course 3, n=20 | 235.95 (93.924)
  Treatment Course 4, n=8: number analyzed (Participants) | 8
  Treatment Course 4, n=8 | 154.88 (19.172)
  Treatment Course 5, n=4: number analyzed (Participants) | 4
  Treatment Course 5, n=4 | 161.75 (22.066)
  Treatment Course 6, n=2: number analyzed (Participants) | 2
  Treatment Course 6, n=2 | 120.00 (0.000)
  Treatment Course 7, n=0: number analyzed (Participants) | 0

5. Secondary Outcome: Ofatumumab Serum Concentration
Description: Blood samples of participants were collected for the measurement of ofatumumab concentration in the blood. The blood samples were collected before infusion (BI) (baseline of that particular treatment course) and at the end of infusion (EI) of ofatumumab.
Time Frame: Before infusion and at the end of infusion for each Treatment Course (8 wk post infusion, then every 4 wk until Wk 24, then every 8 wk until next TC; up to 144 weeks). TCs were individualized based on clinical status and may not correlate to trial vi
Population: FAS Population. Only participants with data available at the particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: Nanograms per milliliter (ng/mL)
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
Nanograms per milliliter (ng/mL)
  Treatment Course 1, Baseline (BI); n=92 | 3596.3 (32324.08)
  Treatment Course 1, Baseline (EI); n=91: number analyzed (Participants) | 91
  Treatment Course 1, Baseline (EI); n=91 | 295588.3 (67754.65)
  Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  Treatment Course 1, Week 104; n=1 | NA (NA) — The mean cannot be calculated for one participant. For this parameter at this time point, the value was below the lower limit of quantification.
  Treatment Course 2, Baseline (BI); n=73: number analyzed (Participants) | 73
  Treatment Course 2, Baseline (BI); n=73 | 837.6 (3102.94)
  Treatment Course 2, Baseline (EI); n=92 | 292283.5 (87672.90)
  Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  Treatment Course 2, Week 80; n=1 | NA (NA) — The mean cannot be calculated for one participant. For this parameter at this time point, the value was below the lower limit of quantification.
  Treatment Course 3, Baseline (BI); n=53: number analyzed (Participants) | 53
  Treatment Course 3, Baseline (BI); n=53 | 955.0 (3270.64)
  Treatment Course 3, Baseline (EI); n=53: number analyzed (Participants) | 53
  Treatment Course 3, Baseline (EI); n=53 | 276719.3 (68620.07)
  Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  Treatment Course 3, Week 64; n=1 | NA (NA) — The mean cannot be calculated for one participant. For this parameter at this time point, the value was below the lower limit of quantification.
  Treatment Course 4, Baseline (BI); n=20: number analyzed (Participants) | 20
  Treatment Course 4, Baseline (BI); n=20 | 2070.2 (3329.24)
  Treatment Course 4, Baseline (EI); n=20: number analyzed (Participants) | 20
  Treatment Course 4, Baseline (EI); n=20 | 296305.7 (76863.21)
  Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  Treatment Course 4, Week 40; n=1 | NA (NA) — The mean cannot be calculated for one participant. For this parameter at this time point, the value was below the lower limit of quantification.
  Treatment Course 5, Baseline (BI); n=8: number analyzed (Participants) | 8
  Treatment Course 5, Baseline (BI); n=8 | 6077.8 (5853.91)
  Treatment Course 5, Baseline (EI); n=8: number analyzed (Participants) | 8
  Treatment Course 5, Baseline (EI); n=8 | 244302.0 (115157.71)
  Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  Treatment Course 5, Week 24; n=2 | 6543.5 (1229.66)
  Treatment Course 6, Baseline (BI); n=4: number analyzed (Participants) | 4
  Treatment Course 6, Baseline (BI); n=4 | 5036.5 (3099.45)
  Treatment Course 6, Baseline (EI); n=4: number analyzed (Participants) | 4
  Treatment Course 6, Baseline (EI); n=4 | 305474.8 (79304.73)
  Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  Treatment Course 6, Week 16; n=2 | 16661.5 (11651.00)
  Treatment Course 7, Baseline (BI); n=2: number analyzed (Participants) | 2
  Treatment Course 7, Baseline (BI); n=2 | 13262.0 (9702.92)
  Treatment Course 7, Baseline (EI); n=2: number analyzed (Participants) | 2
  Treatment Course 7, Baseline (EI); n=2 | 277168.5 (25532.92)
  Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  Treatment Course 7, Week 8; n=2 | 73159.5 (19078.45)

6. Secondary Outcome: Number of Participants Achieving American College of Rheumatology (ACR)20
Description: ACR20 is achieved if the participant has 20% improvement from Baseline in TJC and SJC and in 3 out of 5 of following assessments (A); participant pain A, participant global A, physician global A on a visual analog scale (VAS: a 10 cm scale ranging from "no pain" to "severe pain"; the distance marked by the participant from the "no pain" end is his joint pain score), participant self-assessed disability, and C-reactive protein. The sponsor discontinued the IV administration development program for RA, and this study was terminated early; hence, this endpoint was not evaluated.
Time Frame: Baseline of each TC and 8 wk post infusion, then every 4 wk until Wk 24, then every 8 wk until next treatment course (up to 144 weeks). TCs were individualized based on clinical status and may not correlate to trial visits or study weeks.
Population: FAS Population
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 0

7. Secondary Outcome: Number of Participants Achieving ACR50
Description: ACR50 is achieved if the participant has 50% improvement from Baseline in: TJC and SJC and in 3 out of 5 of following assessment (A) ; participant pain A , participant global A, physician global A on a visual analogue scale (VAS: a 10 cm scale ranges from 'no pain' to 'severe pain' and the distance marked by the participant from the "no pain" end is his joint pain score).and participant self-assessed disability and C-reactive protein. The sponsor discontinued the IV administration development program for RA, and this study was terminated early; hence, this endpoint was not evaluated.
Time Frame: Baseline of each TCand 8 wk post infusion, then every 4 wk until Wk 24, then every 8 wk until next treatment course (up to 144 weeks). TCs were individualized based on clinical status and may not correlate to trial visits or study weeks.
Population: FAS Population
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 0

8. Secondary Outcome: Number of Participants Achieving ACR70
Description: ACR70 is achieved if the participant has 70% improvement from Baseline in: TJC and SJC and in 3 out of 5 of following assessment (A) ; participant pain A , participant global A, physician global A on a visual analogue scale (VAS: a 10 cm scale ranges from 'no pain' to 'severe pain' and the distance marked by the participant from the "no pain" end is his joint pain score).and participant self-assessed disability and C-reactive protein. The sponsor discontinued the IV administration development program for RA, and this study was terminated early; hence, this endpoint was not evaluated.
Time Frame: as for outcome 6
Population: FAS Population
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 0

9. Secondary Outcome: Number of Participants With the Indicated European League Against Rheumatism (EULAR) Response
Description: EULAR response is based on the DAS score. EULAR response criterion classifies participants as good or moderate responders and non-responders. Good response: DAS28 score <=3.2 and >1.2 improvement from Baseline (IfB) in DAS28 score, Moderate response: DAS28 score <=3.2 and between >0.6 and <=1.2 IfB; DAS28 score between >3.2 and <=5.1 and >1.2 IfB; DAS28 score between >3.2 and <=5.1 and between >0.6 and <=1.2 IfB; DAS28 score >5.1 and >1.2 IfB. The sponsor discontinued the IV administration development program for RA, and this study was terminated early; hence, this endpoint was not evaluated.
Time Frame: as for outcome 6
Population: FAS Population
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 0

10. Secondary Outcome: Number of Participants in the Indicated Categories of the Health Assessment Questionnaire (HAQ)
Description: The HAQ, a 20-question instrument, assesses the degree of difficulty a person has in accomplishing tasks in eight functional areas (dressing, arising, eating, walking, hygiene, reaching, gripping, and errands and chores). Responses in each area are scored from 0 (no difficulty) to 3 (inability to perform a task in that area). The index is calculated by adding all scores, then dividing this score by the total number of components answered. The sponsor discontinued the IV administration development program for RA, and this study was terminated early; hence, this endpoint was not evaluated.
Time Frame: as for outcome 6
Population: FAS Population
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 0

11. Secondary Outcome: Number of Participants With the Indicated Global Disease Assessment Using the VAS
Description: The participant and the physician independantly used the VAS for overall assessment of the disease. VAS is used to measure the physician's subjective assessment of the participant's RA disease process at the time of the visit. The scale ranged from 0 (extremely well) to 10 (extremely poor). The sponsor discontinued the IV administration development program for RA, and this study was terminated early; hence, this endpoint was not evaluated.
Time Frame: as for outcome 6
Population: FAS Population
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 0

12. Secondary Outcome: Number of Participants With the Indicated Pain Score
Description: The pain score was assessed using the VAS: a 10 cm scale ranging from "no pain" to "severe pain"; the distance marked by the participant from the "no pain" end is his joint pain score. The sponsor discontinued the IV administration development program for RA, and this study was terminated early; hence, this endpoint was not evaluated.
Time Frame: as for outcome 6
Population: FAS Population
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 0

13. Secondary Outcome: Number of Participants With HAHA Response
Description: The host immune response was assessed based on Human Anti-Human Antibodies (HAHA). The serum samples of the participants were collected for the assessment of HAHA. The sponsor discontinued the IV administration development program for RA, and this study was terminated early; hence, this endpoint was not evaluated.
Time Frame: as for outcome 6
Population: FAS Population
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 0

14. Secondary Outcome: Whole Blood Transcriptional Profiles
Description: Blood samples were collected for transcriptomic analysis of messenger ribonucleic acid (mRNA). The sponsor discontinued the IV administration development program for RA, and this study was terminated early; hence, this endpoint was not evaluated.
Time Frame: as for outcome 6
Population: FAS Population
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 0

15. Secondary Outcome: Percentage of Cluster of Differentiation (CD)19+, 4+, 3+, and 8+ B-cell Subsets in the Blood
Description: Blood samples of participants were collected for the evaluation of CD19+, CD4+, CD3+, and CD8+ B-cell subsets. These biomarkers are associated with immune functions.
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of CD19+, 4+, 8+, and 3+ BCSs
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
Percentage of CD19+, 4+, 8+, and 3+ BCSs
  CD19+, Treatment Course 1, Baseline; n=92 | 6.4 (4.45)
  CD19+, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  CD19+, Treatment Course 1, Week 104; n=1 | 4.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD19+, Treatment Course 2, Baseline; n=72: number analyzed (Participants) | 72
  CD19+, Treatment Course 2, Baseline; n=72 | 1.9 (3.06)
  CD19+, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  CD19+, Treatment Course 2, Week 80; n=1 | 2.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD19+, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  CD19+, Treatment Course 3, Baseline; n=53 | 2.6 (2.99)
  CD19+, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  CD19+, Treatment Course 3, Week 64; n=1 | 1.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD19+, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  CD19+, Treatment Course 4, Baseline; n=20 | 1.7 (2.68)
  CD19+, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  CD19+, Treatment Course 4, Week 40; n=1 | 3.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD19+, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  CD19+, Treatment Course 5, Baseline; n=8 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD19+, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  CD19+, Treatment Course 5, Week 24; n=2 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD19+, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  CD19+, Treatment Course 6, Baseline; n=4 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD19+, Treatment Course 6, Week 12; n=4: number analyzed (Participants) | 4
  CD19+, Treatment Course 6, Week 12; n=4 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD19+, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  CD19+, Treatment Course 7, Baseline; n=2 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD19+, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  CD19+, Treatment Course 7, Week 8; n=2 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD3+, Treatment Course 1, Baseline; n=92 | 79.7 (7.87)
  CD3+, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  CD3+, Treatment Course 1, Week 104; n=1 | 92.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD3+, Treatment Course 2, Baseline; n=72: number analyzed (Participants) | 72
  CD3+, Treatment Course 2, Baseline; n=72 | 81.9 (9.23)
  CD3+, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  CD3+, Treatment Course 2, Week 80; n=1 | 87.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD3+, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  CD3+, Treatment Course 3, Baseline; n=53 | 81.4 (8.84)
  CD3+, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  CD3+, Treatment Course 3, Week 64; n=1 | 77.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD3+, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  CD3+, Treatment Course 4, Baseline; n=20 | 85.4 (5.09)
  CD3+, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  CD3+, Treatment Course 4, Week 40; n=1 | 88.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD3+, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  CD3+, Treatment Course 5, Baseline; n=8 | 86.5 (5.83)
  CD3+, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  CD3+, Treatment Course 5, Week 24; n=2 | 88.5 (0.71)
  CD3+, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  CD3+, Treatment Course 6, Baseline; n=4 | 80.8 (4.57)
  CD3+, Treatment Course 6, Week 12; n=4: number analyzed (Participants) | 4
  CD3+, Treatment Course 6, Week 12; n=4 | 82.8 (5.38)
  CD3+, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  CD3+, Treatment Course 7, Baseline; n=2 | 87.0 (0.00)
  CD3+, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  CD3+, Treatment Course 7, Week 8; n=2 | 84.5 (3.54)
  CD4+, Treatment Course 1, Baseline; n=92 | 51.8 (11.46)
  CD4+, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  CD4+, Treatment Course 1, Week 104; n=1 | 65.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD4+, Treatment Course 2, Baseline; n=72: number analyzed (Participants) | 72
  CD4+, Treatment Course 2, Baseline; n=72 | 53.2 (10.49)
  CD4+, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  CD4+, Treatment Course 2, Week 80; n=1 | 59.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD4+, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  CD4+, Treatment Course 3, Baseline; n=53 | 53.2 (10.72)
  CD4+, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  CD4+, Treatment Course 3, Week 64; n=1 | 58.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD4+, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  CD4+, Treatment Course 4, Baseline; n=20 | 56.6 (13.78)
  CD4+, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  CD4+, Treatment Course 4, Week 40; n=1 | 62.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD4+, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  CD4+, Treatment Course 5, Baseline; n=8 | 53.3 (12.87)
  CD4+, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  CD4+, Treatment Course 5, Week 24; n=2 | 55.5 (17.68)
  CD4+, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  CD4+, Treatment Course 6, Baseline; n=4 | 51.0 (16.06)
  CD4+, Treatment Course 6, Week 12; n=4: number analyzed (Participants) | 4
  CD4+, Treatment Course 6, Week 12; n=4 | 54.8 (17.75)
  CD4+, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  CD4+, Treatment Course 7, Baseline; n=2 | 57.0 (9.90)
  CD4+, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  CD4+, Treatment Course 7, Week 8; n=2 | 54.5 (16.26)
  CD8+, Treatment Course 1, Baseline; n=92 | 23.7 (8.61)
  CD8+, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  CD8+, Treatment Course 1, Week 104; n=1 | 23.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD8+, Treatment Course 2, Baseline; n=72: number analyzed (Participants) | 72
  CD8+, Treatment Course 2, Baseline; n=72 | 24.2 (7.94)
  CD8+, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  CD8+, Treatment Course 2, Week 80; n=1 | 26.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD8+, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  CD8+, Treatment Course 3, Baseline; n=53 | 24.1 (7.83)
  CD8+, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  CD8+, Treatment Course 3, Week 64; n=1 | 18.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD8+, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  CD8+, Treatment Course 4, Baseline; n=20 | 24.6 (8.24)
  CD8+, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  CD8+, Treatment Course 4, Week 40; n=1 | 22.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD8+, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  CD8+, Treatment Course 5, Baseline; n=8 | 27.5 (9.47)
  CD8+, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  CD8+, Treatment Course 5, Week 24; n=2 | 23.5 (7.78)
  CD8+, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  CD8+, Treatment Course 6, Baseline; n=4 | 26.0 (10.10)
  CD8+, Treatment Course 6, Week 12; n=4: number analyzed (Participants) | 4
  CD8+, Treatment Course 6, Week 12; n=4 | 24.3 (11.15)
  CD8+, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  CD8+, Treatment Course 7, Baseline; n=2 | 26.0 (8.49)
  CD8+, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  CD8+, Treatment Course 7, Week 8; n=2 | 25.5 (10.61)

16. Secondary Outcome: CD19+, CD4+, CD3+, and CD8+ Cell Counts, Measured in mm^3
Description: Blood samples of participants were collected for the evaluation of CD19+, CD4+, CD3+, and CD8+ cell counts. These cells are present on white blood cells and are used as markers to associate cells with immune functions.
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: cells per millimeters cubed (mm^3)
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
cells per millimeters cubed (mm^3)
  CD19+, Treatment Course 1, Baseline; n=92 | 109.6 (91.12)
  CD19+, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  CD19+, Treatment Course 1, Week 104; n=1 | 95.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD19+, Treatment Course 2, Baseline; n=71: number analyzed (Participants) | 71
  CD19+, Treatment Course 2, Baseline; n=71 | 30.0 (49.36)
  CD19+, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  CD19+, Treatment Course 2, Week 80; n=1 | 24.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD19+, Treatment Course 3, Baseline; n=51: number analyzed (Participants) | 51
  CD19+, Treatment Course 3, Baseline; n=51 | 43.8 (50.11)
  CD19+, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  CD19+, Treatment Course 3, Week 64; n=1 | 16.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD19+, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  CD19+, Treatment Course 4, Baseline; n=20 | 27.2 (43.75)
  CD19+, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  CD19+, Treatment Course 4, Week 40; n=1 | 54.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD19+, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  CD19+, Treatment Course 5, Baseline; n=8 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD19+, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  CD19+, Treatment Course 5, Week 24; n=2 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD19+, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  CD19+, Treatment Course 6, Baseline; n=4 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD19+, Treatment Course 6, Week 12; n=4: number analyzed (Participants) | 4
  CD19+, Treatment Course 6, Week 12; n=4 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD19+, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  CD19+, Treatment Course 7, Baseline; n=2 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD19+, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  CD19+, Treatment Course 7, Week 8; n=2 | 0 (NA) — A dispersion cannot be calculated for a mean of 0.
  CD3+, Treatment Course 1, Baseline; n=92 | 1325.3 (467.40)
  CD3+, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  CD3+, Treatment Course 1, Week 104; n=1 | 2174.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CD3+, Treatment Course 2, Baseline; n=71: number analyzed (Participants) | 71
  CD3+, Treatment Course 2, Baseline; n=71 | 1338.8 (557.04)
  CD3+, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  CD3+, Treatment Course 2, Week 80; n=1 | 1051.0 (NA) — Standard deviation is not calculated when only one participant was analyzed
  CD3+, Treatment Course 3, Baseline; n=51: number analyzed (Participants) | 51
  CD3+, Treatment Course 3, Baseline; n=51 | 1325.1 (398.74)
  CD3+, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  CD3+, Treatment Course 3, Week 64; n=1 | 1213.0 (NA) — Standard deviation is not calculated when only one participant was analyzed
  CD3+, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  CD3+, Treatment Course 4, Baseline; n=20 | 1388.3 (502.80)
  CD3+, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  CD3+, Treatment Course 4, Week 40; n=1 | 1594.0 (NA) — Standard deviation is not calculated when only one participant was analyzed
  CD3+, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  CD3+, Treatment Course 5, Baseline; n=8 | 1324.1 (618.65)
  CD3+, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  CD3+, Treatment Course 5, Week 24; n=2 | 1218.5 (342.95)
  CD3+, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  CD3+, Treatment Course 6, Baseline; n=4 | 1574.3 (553.71)
  CD3+, Treatment Course 6, Week 12; n=4: number analyzed (Participants) | 4
  CD3+, Treatment Course 6, Week 12; n=4 | 1430.8 (507.31)
  CD3+, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  CD3+, Treatment Course 7, Baseline; n=2 | 1062.0 (169.71)
  CD3+, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  CD3+, Treatment Course 7, Week 8; n=2 | 1230.0 (373.35)
  CD4+, Treatment Course 1, Baseline; n=92 | 869.2 (386.45)
  CD4+, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  CD4+, Treatment Course 1, Week 104; n=1 | 1544.0 (NA) — Standard deviation is not calculated when only one participant was analyzed
  CD4+, Treatment Course 2, Baseline; n=71: number analyzed (Participants) | 71
  CD4+, Treatment Course 2, Baseline; n=71 | 877.3 (443.09)
  CD4+, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  CD4+, Treatment Course 2, Week 80; n=1 | 715.0 (NA) — Standard deviation is not calculated when only one participant was analyzed
  CD4+, Treatment Course 3, Baseline; n=51: number analyzed (Participants) | 51
  CD4+, Treatment Course 3, Baseline; n=51 | 876.7 (310.96)
  CD4+, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  CD4+, Treatment Course 3, Week 64; n=1 | 910.0 (NA) — Standard deviation is not calculated when only one participant was analyzed
  CD4+, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  CD4+, Treatment Course 4, Baseline; n=20 | 931.8 (451.30)
  CD4+, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  CD4+, Treatment Course 4, Week 40; n=1 | 1116.0 (NA) — Standard deviation is not calculated when only one participant was analyzed
  CD4+, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  CD4+, Treatment Course 5, Baseline; n=8 | 837.3 (499.45)
  CD4+, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  CD4+, Treatment Course 5, Week 24; n=2 | 729.0 (18.38)
  CD4+, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  CD4+, Treatment Course 6, Baseline; n=4 | 1000.3 (545.33)
  CD4+, Treatment Course 6, Week 12; n=4: number analyzed (Participants) | 4
  CD4+, Treatment Course 6, Week 12; n=4 | 919.8 (380.08)
  CD4+, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  CD4+, Treatment Course 7, Baseline; n=2 | 686.0 (1.41)
  CD4+, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  CD4+, Treatment Course 7, Week 8; n=2 | 755.5 (30.41)
  CD8+, Treatment Course 1, Baseline; n=92 | 387.7 (183.18)
  CD8+, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  CD8+, Treatment Course 1, Week 104; n=1 | 543.0 (NA) — Standard deviation is not calculated when only one participant was analyzed
  CD8+, Treatment Course 2, Baseline; n=71: number analyzed (Participants) | 71
  CD8+, Treatment Course 2, Baseline; n=71 | 391.0 (193.89)
  CD8+, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  CD8+, Treatment Course 2, Week 80; n=1 | 315.0 (NA) — Standard deviation is not calculated when only one participant was analyzed
  CD8+, Treatment Course 3, Baseline; n=51: number analyzed (Participants) | 51
  CD8+, Treatment Course 3, Baseline; n=51 | 383.3 (159.28)
  CD8+, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  CD8+, Treatment Course 3, Week 64; n=1 | 279.0 (NA) — Standard deviation is not calculated when only one participant was analyzed
  CD8+, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  CD8+, Treatment Course 4, Baseline; n=20 | 389.0 (151.22)
  CD8+, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  CD8+, Treatment Course 4, Week 40; n=1 | 398.0 (NA) — Standard deviation is not calculated when only one participant was analyzed
  CD8+, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  CD8+, Treatment Course 5, Baseline; n=8 | 411.0 (198.41)
  CD8+, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  CD8+, Treatment Course 5, Week 24; n=2 | 338.5 (202.94)
  CD8+, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  CD8+, Treatment Course 6, Baseline; n=4 | 502.3 (234.80)
  CD8+, Treatment Course 6, Week 12; n=4: number analyzed (Participants) | 4
  CD8+, Treatment Course 6, Week 12; n=4 | 443.8 (298.72)
  CD8+, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  CD8+, Treatment Course 7, Baseline; n=2 | 327.0 (155.56)
  CD8+, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  CD8+, Treatment Course 7, Week 8; n=2 | 400.0 (278.60)

17. Secondary Outcome: Ratio of CD 4+/CD8+
Description: Blood samples of participants were collected for the evaluation of CD4+ and CD8+ cell counts and the ratio was calculated.
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: Ratio of CD 4+/CD8+ cells
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 72
Ratio of CD 4+/CD8+ cells
  Treatment Course 1, Baseline; n=72 | 2.55 (1.295)
  Treatment Course 1, Week 48; n=1: number analyzed (Participants) | 1
  Treatment Course 1, Week 48; n=1 | 5.40 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Treatment Course 2, Week 24; n=1: number analyzed (Participants) | 1
  Treatment Course 2, Week 24; n=1 | 4.10 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Treatment Course 2, Week 56; n=1: number analyzed (Participants) | 1
  Treatment Course 2, Week 56; n=1 | 2.60 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Treatment Course 3, Baseline; n=1: number analyzed (Participants) | 1
  Treatment Course 3, Baseline; n=1 | 2.60 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Treatment Course 3, Week 32; n=2: number analyzed (Participants) | 2
  Treatment Course 3, Week 32; n=2 | 2.40 (0.424)
  Treatment Course 4, Baseline; n=1: number analyzed (Participants) | 1
  Treatment Course 4, Baseline; n=1 | 1.50 (NA) — Standard deviation is not calculated when only one participant was analyzed.

18. Secondary Outcome: Number of Participants With Rheumatoid Factor (RA Factor) >13 International Units Per Milliliter
Description: Blood samples of participants were collected for the evaulation of RA factor. RA factor is an antibody found in the blood of participants with rheumatoid arthritis and is used for the diagnosis of rheumatoid arthritis.
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
participants
  Treatment Course 1, Baseline; n=92 | 79
  Treatment Course 1, Week 104; n=1 | 1
  Treatment Course 1, At any time; n=92 | 81
  Treatment Course 2, Baseline; n=73 | 60
  Treatment Course 2, Week 80; n=1 | 1
  Treatment Course 2, At any time; n=73 | 63
  Treatment Course 3, Baseline; n=53 | 42
  Treatment Course 3, Week 64; n=1 | 1
  Treatment Course 3, At any time; n=53 | 46
  Treatment Course 4, Baseline; n=20 | 13
  Treatment Course 4, Week 40; n=1 | 1
  Treatment Course 4, At any time; n=20 | 14
  Treatment Course 5, Baseline; n=8 | 4
  Treatment Course 5, Week 24; n=2 | 0
  Treatment Course 5, At any time; n=8 | 4
  Treatment Course 6, Baseline; n=4 | 2
  Treatment Course 6, Week 16; n=2 | 1
  Treatment Course 6, At any time; n=4 | 2
  Treatment Course 7, Baseline; n=2 | 1
  Treatment Course 7, Week 8; n=2 | 1
  Treatment Course 7, At any time; n=2 | 1

19. Secondary Outcome: Number of Participants With Anti-cyclic Citrullinated Peptide Antibody (CCP) >6.9 International Units Per Liter
Description: Blood samples of participants were collected for the evaluation of Anti-CCP. Anti-CCP plays an important role in immune response and helps assess the disease condition.
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
participants
  Treatment Course 1, Baseline; n=92 | 80
  Treatment Course 1, Week 104; n=1 | 1
  Treatment Course 1, At any time; n=92 | 83
  Treatment Course 2, Baseline; n=73 | 66
  Treatment Course 2, Week 80; n=1 | 1
  Treatment Course 2, At any time; n=73 | 67
  Treatment Course 3, Baseline; n=53 | 48
  Treatment Course 3, Week 64; n=1 | 1
  Treatment Course 3, At any time; n=53 | 48
  Treatment Course 4, Baseline; n=20 | 15
  Treatment Course 4, Week 40; n=1 | 1
  Treatment Course 4, At any time; n=20 | 15
  Treatment Course 5, Baseline; n=8 | 7
  Treatment Course 5, Week 24; n=2 | 1
  Treatment Course 5, At any time; n=8 | 7
  Treatment Course 6, Baseline; n=4 | 3
  Treatment Course 6, Week 16; n=2 | 1
  Treatment Course 6, At any time; n=4 | 3
  Treatment Course 7, Baseline; n=2 | 1
  Treatment Course 7, Week 8; n=2 | 1
  Treatment Course 7, At any time; n=2 | 1

20. Secondary Outcome: Number of Participants With B-Lymphocyte Stimulator (BLyS) >2.49 Micrograms Per Liter
Description: Blood samples of participants were collected for the evaluation of BLyS. BLyS is a potent co-stimulator of B lymphocytes, and elevated levels of BLyS are observed in automimmune diseases. It regulates the immunnoglobin (antibody produced by B cells that is used by the immune system to indentify bacteria and viruses in the body) secretion of normal B cells (type of cells in the blood).
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
participants
  Treatment Course 1, Baseline; n=92 | 12
  Treatment Course 1, Week 104; n=1 | 0
  Treatment Course 1, At any time; n=92 | 81
  Treatment Course 2, Baseline; n=73 | 38
  Treatment Course 2, Week 80; n=1 | 0
  Treatment Course 2, At any time; n=73 | 65
  Treatment Course 3, Baseline; n=53 | 32
  Treatment Course 3, Week 64; n=1 | 1
  Treatment Course 3, At any time; n=53 | 48
  Treatment Course 4, Baseline; n=20 | 12
  Treatment Course 4, Week 40; n=1 | 1
  Treatment Course 4, At any time; n=20 | 16
  Treatment Course 5, Baseline; n=8 | 7
  Treatment Course 5, Week 24; n=2 | 2
  Treatment Course 5, At any time; n=8 | 7
  Treatment Course 6, Baseline; n=4 | 4
  Treatment Course 6, Week 16; n=2 | 2
  Treatment Course 6, At any time; n=4 | 4
  Treatment Course 7, Baseline; n=2 | 2
  Treatment Course 7, Week 8; n=2 | 2
  Treatment Course 7, At any time; n=2 | 2

21. Secondary Outcome: Number of Participants With Interleukin 6 (IL-6) >11.9 Picograms Per Milliliter
Description: Blood samples of participants were collected for the evaluation of IL-6. IL-6 plays an important role in immune response and helps assess the disease condition.
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
participants
  Treatment Course 1, Baseline; n=92 | 40
  Treatment Course 1, Week 104; n=1 | 0
  Treatment Course 1, At any time; n=92 | 47
  Treatment Course 2, Baseline; n=73 | 12
  Treatment Course 2, Week 80; n=1 | 1
  Treatment Course 2, At any time; n=73 | 27
  Treatment Course 3, Baseline; n=52 | 11
  Treatment Course 3, Week 64; n=1 | 0
  Treatment Course 3, At any time; n=53 | 15
  Treatment Course 4, Baseline; n=20 | 3
  Treatment Course 4, Week 40; n=1 | 0
  Treatment Course 4, At any time; n=20 | 4
  Treatment Course 5, Baseline; n=8 | 1
  Treatment Course 5, Week 24; n=2 | 0
  Treatment Course 5, At any time; n=8 | 1
  Treatment Course 6, Baseline; n=4 | 0
  Treatment Course 6, Week 16; n=2 | 0
  Treatment Course 6, At any time; n=4 | 0
  Treatment Course 7, Baseline; n=2 | 0
  Treatment Course 7, Week 8; n=2 | 0
  Treatment Course 7, At any time; n=2 | 0

22. Secondary Outcome: Assessment of Sodium, Potassium, Chloride, Bicarbonate, Calcium, and Uric Acid
Description: Blood samples of participants were collected for the evaluation of uric acid and electrolytes (sodium, potassium, chloride, and calcium), as increased levels may reflect B-cell lysis due to treatment with ofatumumab.
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimoles/liter (mmol/L)
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
Millimoles/liter (mmol/L)
  Sodium, Treatment Course 1, Baseline; n=92 | 142.1 (2.76)
  Sodium, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  Sodium, Treatment Course 1, Week 104; n=1 | 144.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Sodium, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  Sodium, Treatment Course 2, Baseline; n=73 | 142.3 (2.25)
  Sodium, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  Sodium, Treatment Course 2, Week 80; n=1 | 145.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Sodium, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  Sodium, Treatment Course 3, Baseline; n=53 | 143.3 (2.26)
  Sodium, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  Sodium, Treatment Course 3, Week 64; n=1 | 147.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Sodium, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  Sodium, Treatment Course 4, Baseline; n=20 | 142.8 (2.65)
  Sodium, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  Sodium, Treatment Course 4, Week 40; n=1 | 145.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Sodium, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  Sodium, Treatment Course 5, Baseline; n=8 | 143.1 (2.30)
  Sodium, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  Sodium, Treatment Course 5, Week 24; n=2 | 142.5 (2.12)
  Sodium, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  Sodium, Treatment Course 6, Baseline; n=4 | 142.0 (1.83)
  Sodium, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  Sodium, Treatment Course 6, Week 16; n=2 | 141.5 (3.54)
  Sodium, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  Sodium, Treatment Course 7, Baseline; n=2 | 142.5 (0.71)
  Sodium, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  Sodium, Treatment Course 7, Week 8; n=2 | 141.0 (2.83)
  Potassium, Treatment Course 1, Baseline; n=92 | 4.25 (0.317)
  Potassium, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  Potassium, Treatment Course 1, Week 104; n=1 | 3.30 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Potassium, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  Potassium, Treatment Course 2, Baseline; n=73 | 4.32 (0.386)
  Potassium, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  Potassium, Treatment Course 2, Week 80; n=1 | 4.20 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Potassium, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  Potassium, Treatment Course 3, Baseline; n=53 | 4.25 (0.358)
  Potassium, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  Potassium, Treatment Course 3, Week 64; n=1 | 4.60 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Potassium, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  Potassium, Treatment Course 4, Baseline; n=20 | 4.20 (0.208)
  Potassium, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  Potassium, Treatment Course 4, Week 40; n=1 | 4.20 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Potassium, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  Potassium, Treatment Course 5, Baseline; n=8 | 4.34 (0.220)
  Potassium, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  Potassium, Treatment Course 5, Week 24; n=2 | 4.40 (0.283)
  Potassium, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  Potassium, Treatment Course 6, Baseline; n=4 | 4.48 (0.377)
  Potassium, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  Potassium, Treatment Course 6, Week 16; n=2 | 4.45 (0.495)
  Potassium, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  Potassium, Treatment Course 7, Baseline; n=2 | 4.50 (0.707)
  Potassium, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  Potassium, Treatment Course 7, Week 8; n=2 | 4.35 (0.495)
  Chloride, Treatment Course 1, Baseline; n=92 | 105.2 (2.98)
  Chloride, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  Chloride, Treatment Course 1, Week 104; n=1 | 104.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Chloride Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  Chloride Treatment Course 2, Baseline; n=73 | 105.6 (2.18)
  Chloride Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  Chloride Treatment Course 2, Week 80; n=1 | 105.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Chloride, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  Chloride, Treatment Course 3, Baseline; n=53 | 106.0 (2.54)
  Chloride, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  Chloride, Treatment Course 3, Week 64; n=1 | 111.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Chloride Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  Chloride Treatment Course 4, Baseline; n=20 | 105.9 (3.56)
  Chloride, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  Chloride, Treatment Course 4, Week 40; n=1 | 102.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Chloride Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  Chloride Treatment Course 5, Baseline; n=8 | 104.8 (3.54)
  Chloride, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  Chloride, Treatment Course 5, Week 24; n=2 | 105.5 (3.54)
  Chloride, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  Chloride, Treatment Course 6, Baseline; n=4 | 105.0 (3.37)
  Chloride, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  Chloride, Treatment Course 6, Week 16; n=2 | 105.0 (2.83)
  Chloride, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  Chloride, Treatment Course 7, Baseline; n=2 | 104.0 (1.41)
  Chloride, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  Chloride, Treatment Course 7, Week 8; n=2 | 105.0 (4.24)
  Bicarbonate, Treatment Course 1, Baseline; n=92 | 24.67 (2.519)
  Bicarbonate, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  Bicarbonate, Treatment Course 1, Week 104; n=1 | 28.40 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Bicarbonate, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  Bicarbonate, Treatment Course 2, Baseline; n=73 | 25.10 (2.416)
  Bicarbonate, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  Bicarbonate, Treatment Course 2, Week 80; n=1 | 22.80 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Bicarbonate, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  Bicarbonate, Treatment Course 3, Baseline; n=53 | 25.49 (2.299)
  Bicarbonate, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  Bicarbonate, Treatment Course 3, Week 64; n=1 | 25.40 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Bicarbonate, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  Bicarbonate, Treatment Course 4, Baseline; n=20 | 24.61 (2.748)
  Bicarbonate, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  Bicarbonate, Treatment Course 4, Week 40; n=1 | 30.00 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Bicarbonate, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  Bicarbonate, Treatment Course 5, Baseline; n=8 | 26.20 (2.262)
  Bicarbonate, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  Bicarbonate, Treatment Course 5, Week 24; n=2 | 27.20 (4.243)
  Bicarbonate, , Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  Bicarbonate, , Treatment Course 6, Baseline; n=4 | 25.00 (0.876)
  Bicarbonate, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  Bicarbonate, Treatment Course 6, Week 16; n=2 | 24.50 (2.546)
  Bicarbonate, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  Bicarbonate, Treatment Course 7, Baseline; n=2 | 24.80 (1.414)
  Bicarbonate, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  Bicarbonate, Treatment Course 7, Week 8; n=2 | 23.40 (0.849)
  Calcium, Treatment Course 1, Baseline; n=92 | 2.324 (0.0965)
  Calcium Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  Calcium Treatment Course 1, Week 104; n=1 | 2.250 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Calcium, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  Calcium, Treatment Course 2, Baseline; n=73 | 2.305 (0.0991)
  Calcium, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  Calcium, Treatment Course 2, Week 80; n=1 | 2.200 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Calcium, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  Calcium, Treatment Course 3, Baseline; n=53 | 2.312 (0.0935)
  Calcium, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  Calcium, Treatment Course 3, Week 64; n=1 | 2.300 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Calcium, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  Calcium, Treatment Course 4, Baseline; n=20 | 2.315 (0.1113)
  Calcium, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  Calcium, Treatment Course 4, Week 40; n=1 | 2.400 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Calcium, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  Calcium, Treatment Course 5, Baseline; n=8 | 2.313 (0.0954)
  Calcium, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  Calcium, Treatment Course 5, Week 24; n=2 | 2.275 (0.1061)
  Calcium, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  Calcium, Treatment Course 6, Baseline; n=4 | 2.338 (0.1109)
  Calcium, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  Calcium, Treatment Course 6, Week 16; n=2 | 2.275 (0.1061)
  Calcium, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  Calcium, Treatment Course 7, Baseline; n=2 | 2.375 (0.1768)
  Calcium, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  Calcium, Treatment Course 7, Week 8; n=2 | 2.300 (0.0707)
  Uric acid, Treatment Course 1, Baseline; n=92 | 0.259 (0.0684)
  Uric acid, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  Uric acid, Treatment Course 1, Week 104; n=1 | 0.380 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Uric acid, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  Uric acid, Treatment Course 2, Baseline; n=73 | 0.265 (0.0572)
  Uric acid, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  Uric acid, Treatment Course 2, Week 80; n=1 | 0.300 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Uric acid, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  Uric acid, Treatment Course 3, Baseline; n=53 | 0.259 (0.0502)
  Uric acid, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  Uric acid, Treatment Course 3, Week 64; n=1 | 0.250 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Uric acid, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  Uric acid, Treatment Course 4, Baseline; n=20 | 0.256 (0.0518)
  Uric acid, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  Uric acid, Treatment Course 4, Week 40; n=1 | 0.310 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Uric acid, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  Uric acid, Treatment Course 5, Baseline; n=8 | 0.275 (0.0407)
  Uric acid, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  Uric acid, Treatment Course 5, Week 24; n=2 | 0.245 (0.0354)
  Uric acid, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  Uric acid, Treatment Course 6, Baseline; n=4 | 0.273 (0.0222)
  Uric acid, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  Uric acid, Treatment Course 6, Week 16; n=2 | 0.265 (0.0212)
  Uric acid, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  Uric acid, Treatment Course 7, Baseline; n=2 | 0.250 (0.0424)
  Uric acid, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  Uric acid, Treatment Course 7, Week 8; n=2 | 0.295 (0.0354)

23. Secondary Outcome: Assessment of Total Protein (TP) and Albumin
Description: Blood samples of participants were collected to evaluate TP and albumin. TP can vary depending on auto-immune diseases, and TP and albumin can vary depending on debilitating diseases.
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: Grams/Liter (g/L)
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
Grams/Liter (g/L)
  TP, Treatment Course 1, Baseline; n=92 | 76.3 (4.97)
  TP, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  TP, Treatment Course 1, Week 104; n=1 | 72.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  TP, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  TP, Treatment Course 2, Baseline; n=73 | 76.2 (4.53)
  TP, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  TP, Treatment Course 2, Week 80; n=1 | 72.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  TP, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  TP, Treatment Course 3, Baseline; n=53 | 74.7 (4.80)
  TP, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  TP, Treatment Course 3, Week 64; n=1 | 71.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  TP, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  TP, Treatment Course 4, Baseline; n=20 | 73.9 (5.44)
  TP, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  TP, Treatment Course 4, Week 40; n=1 | 78.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  TP, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  TP, Treatment Course 5, Baseline; n=8 | 75.6 (4.17)
  TP, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  TP, Treatment Course 5, Week 24; n=2 | 75.0 (5.66)
  TP, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  TP, Treatment Course 6, Baseline; n=4 | 74.8 (4.50)
  TP, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  TP, Treatment Course 6, Week 16; n=2 | 77.0 (5.66)
  TP, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  TP, Treatment Course 7, Baseline; n=2 | 78.5 (6.36)
  TP, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  TP, Treatment Course 7, Week 8; n=2 | 75.0 (2.83)
  Albumin, Treatment Course 1, Baseline; n=92 | 43.50 (3.043)
  Albumin, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  Albumin, Treatment Course 1, Week 104; n=1 | 40.80 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Albumin, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  Albumin, Treatment Course 2, Baseline; n=73 | 44.21 (2.984)
  Albumin, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  Albumin, Treatment Course 2, Week 80; n=1 | 39.10 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Albumin, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  Albumin, Treatment Course 3, Baseline; n=53 | 44.18 (3.332)
  Albumin, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  Albumin, Treatment Course 3, Week 64; n=1 | 43.40 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Albumin, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  Albumin, Treatment Course 4, Baseline; n=20 | 44.34 (3.497)
  Albumin, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  Albumin, Treatment Course 4, Week 40; n=1 | 46.20 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Albumin, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  Albumin, Treatment Course 5, Baseline; n=8 | 46.75 (3.203)
  Albumin, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  Albumin, Treatment Course 5, Week 24; n=2 | 45.90 (2.263)
  Albumin, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  Albumin, Treatment Course 6, Baseline; n=4 | 45.83 (3.035)
  Albumin, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  Albumin, Treatment Course 6, Week 16; n=2 | 46.80 (2.546)
  Albumin, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  Albumin, Treatment Course 7, Baseline; n=2 | 48.00 (3.536)
  Albumin, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  Albumin, Treatment Course 7, Week 8; n=2 | 45.75 (1.344)
  Albumin, Follow-up Week 12; n=59: number analyzed (Participants) | 59
  Albumin, Follow-up Week 12; n=59 | 43.93 (3.002)
  Albumin, Follow-up Week 24; n=18: number analyzed (Participants) | 18
  Albumin, Follow-up Week 24; n=18 | 44.66 (3.642)

24. Secondary Outcome: Assessment of Total Bilirubin (TB) and Creatinine
Description: Blood samples of participants were collected to evaluatate TB and creatinine levles. TB evlauation is performed to assess the condition of the liver, and possible hemolytic anemia, and the creatinine evaulation is performed to assess the renal condition (condition of the kidneys).
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: Micromoles per liter (umol/L)
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
Micromoles per liter (umol/L)
  TB, Treatment Course 1, Baseline; n=92 | 7.18 (3.823)
  TB, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  TB, Treatment Course 1, Week 104; n=1 | 6.30 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  TB, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  TB, Treatment Course 2, Baseline; n=73 | 7.91 (4.528)
  TB, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  TB, Treatment Course 2, Week 80; n=1 | 3.10 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  TB, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  TB, Treatment Course 3, Baseline; n=53 | 7.84 (4.501)
  TB, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  TB, Treatment Course 3, Week 64; n=1 | 8.00 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  TB, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  TB, Treatment Course 4, Baseline; n=20 | 7.68 (3.652)
  TB, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  TB, Treatment Course 4, Week 40; n=1 | 7.50 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  TB, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  TB, Treatment Course 5, Baseline; n=8 | 9.20 (5.283)
  TB, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  TB, Treatment Course 5, Week 24; n=2 | 6.40 (2.546)
  TB, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  TB, Treatment Course 6, Baseline; n=4 | 10.38 (3.779)
  TB, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  TB, Treatment Course 6, Week 16; n=2 | 9.85 (0.636)
  TB, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  TB, Treatment Course 7, Baseline; n=2 | 8.95 (1.344)
  TB, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  TB, Treatment Course 7, Week 8; n=2 | 14.05 (5.586)
  Creatinine, Treatment Course 1, Baseline; n=92 | 64.14 (12.569)
  Creatinine, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  Creatinine, Treatment Course 1, Week 104; n=1 | 54.80 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Creatinine, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  Creatinine, Treatment Course 2, Baseline; n=73 | 67.82 (14.735)
  Creatinine, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  Creatinine, Treatment Course 2, Week 80; n=1 | 75.10 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Creatinine, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  Creatinine, Treatment Course 3, Baseline; n=53 | 65.50 (10.871)
  Creatinine, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  Creatinine, Treatment Course 3, Week 64; n=1 | 68.10 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Creatinine, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  Creatinine, Treatment Course 4, Baseline; n=20 | 65.36 (12.626)
  Creatinine, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  Creatinine, Treatment Course 4, Week 40; n=1 | 70.70 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Creatinine, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  Creatinine, Treatment Course 5, Baseline; n=8 | 67.75 (7.543)
  Creatinine, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  Creatinine, Treatment Course 5, Week 24; n=2 | 64.55 (6.293)
  Creatinine, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  Creatinine, Treatment Course 6, Baseline; n=4 | 67.63 (11.909)
  Creatinine, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  Creatinine, Treatment Course 6, Week 16; n=2 | 60.55 (8.132)
  Creatinine, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  Creatinine, Treatment Course 7, Baseline; n=2 | 61.40 (13.111)
  Creatinine, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  Creatinine, Treatment Course 7, Week 8; n=2 | 59.65 (9.405)
  Creatinine, Follow-up Week 12; n=59: number analyzed (Participants) | 59
  Creatinine, Follow-up Week 12; n=59 | 69.72 (15.553)
  Creatinine, Follow-up Week 24; n=18: number analyzed (Participants) | 18
  Creatinine, Follow-up Week 24; n=18 | 74.95 (21.833)

25. Secondary Outcome: Assessment of Alanine Aminotranferase (ALT), Aspartate Aminotransferase (AST), Alkaline Phosphatase (AP), and Gamma Glutamyl-transferase (GGT)
Description: Blood samples of participants were collected for the evaluation of ALT, AST, AP, and GGT. AST, ALT, AP, and GGT are evaluated to assess the condition of the liver.
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: Units per liter (U/L)
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
Units per liter (U/L)
  ALT, Treatment Course 1, Baseline; n=92 | 20.4 (11.71)
  ALT, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  ALT, Treatment Course 1, Week 104; n=1 | 16.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  ALT, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  ALT, Treatment Course 2, Baseline; n=73 | 21.8 (11.99)
  ALT, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  ALT, Treatment Course 2, Week 80; n=1 | 19.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  ALT, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  ALT, Treatment Course 3, Baseline; n=53 | 20.5 (15.40)
  ALT, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  ALT, Treatment Course 3, Week 64; n=1 | 36.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  ALT, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  ALT, Treatment Course 4, Baseline; n=20 | 22.7 (12.39)
  ALT, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  ALT, Treatment Course 4, Week 40; n=1 | 19.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  ALT, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  ALT, Treatment Course 5, Baseline; n=8 | 19.0 (5.04)
  ALT, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  ALT, Treatment Course 5, Week 24; n=2 | 15.0 (1.41)
  ALT, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  ALT, Treatment Course 6, Baseline; n=4 | 23.5 (9.43)
  ALT, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  ALT, Treatment Course 6, Week 16; n=2 | 24.0 (1.41)
  ALT, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  ALT, Treatment Course 7, Baseline; n=2 | 18.5 (2.12)
  ALT, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  ALT, Treatment Course 7, Week 8; n=2 | 22.0 (4.24)
  AST, Treatment Course 1, Baseline; n=92 | 21.1 (9.01)
  AST, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  AST, Treatment Course 1, Week 104; n=1 | 17.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  AST, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  AST, Treatment Course 2, Baseline; n=73 | 22.8 (8.96)
  AST, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  AST, Treatment Course 2, Week 80; n=1 | 21.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  AST, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  AST, Treatment Course 3, Baseline; n=53 | 21.8 (10.83)
  AST, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  AST, Treatment Course 3, Week 64; n=1 | 21.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  AST, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  AST, Treatment Course 4, Baseline; n=20 | 21.2 (6.47)
  AST, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  AST, Treatment Course 4, Week 40; n=1 | 23.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  AST, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  AST, Treatment Course 5, Baseline; n=8 | 22.4 (7.78)
  AST, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  AST, Treatment Course 5, Week 24; n=2 | 18.0 (0.00)
  AST, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  AST, Treatment Course 6, Baseline; n=4 | 25.3 (8.77)
  AST, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  AST, Treatment Course 6, Week 16; n=2 | 23.5 (3.54)
  AST, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  AST, Treatment Course 7, Baseline; n=2 | 22.5 (4.95)
  AST, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  AST, Treatment Course 7, Week 8; n=2 | 21.5 (0.71)
  AP, Treatment Course 1, Baseline; n=92 | 79.4 (27.80)
  AP, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  AP, Treatment Course 1, Week 104; n=1 | 60.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  AP, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  AP, Treatment Course 2, Baseline; n=73 | 73.3 (23.76)
  AP, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  AP, Treatment Course 2, Week 80; n=1 | 79.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  AP, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  AP, Treatment Course 3, Baseline; n=53 | 70.5 (22.18)
  AP, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  AP, Treatment Course 3, Week 64; n=1 | 61.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  AP, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  AP, Treatment Course 4, Baseline; n=20 | 66.2 (15.54)
  AP, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  AP, Treatment Course 4, Week 40; n=1 | 77.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  AP, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  AP, Treatment Course 5, Baseline; n=8 | 68.0 (25.03)
  AP, Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  AP, Treatment Course 5, Week 24; n=2 | 52.0 (14.14)
  AP, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  AP, Treatment Course 6, Baseline; n=4 | 59.5 (26.51)
  AP, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  AP, Treatment Course 6, Week 16; n=2 | 49.0 (1.41)
  AP, Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  AP, Treatment Course 7, Baseline; n=2 | 47.5 (2.12)
  AP, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  AP, Treatment Course 7, Week 8; n=2 | 45.0 (2.83)
  GGT, Treatment Course 1, Baseline; n=92 | 22.2 (18.51)
  GGT, Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  GGT, Treatment Course 1, Week 104; n=1 | 16.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  GGT, Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  GGT, Treatment Course 2, Baseline; n=73 | 22.0 (20.88)
  GGT, Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  GGT, Treatment Course 2, Week 80; n=1 | 21.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  GGT, Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  GGT, Treatment Course 3, Baseline; n=53 | 19.0 (12.78)
  GGT, Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  GGT, Treatment Course 3, Week 64; n=1 | 50.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  GGT, Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  GGT, Treatment Course 4, Baseline; n=20 | 16.4 (8.41)
  GGT, Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  GGT, Treatment Course 4, Week 40; n=1 | 12.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  GGT, Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  GGT, Treatment Course 5, Baseline; n=8 | 14.4 (2.97)
  GGT Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  GGT Treatment Course 5, Week 24; n=2 | 11.0 (1.41)
  GGT, Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  GGT, Treatment Course 6, Baseline; n=4 | 16.5 (7.19)
  GGT, Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  GGT, Treatment Course 6, Week 16; n=2 | 14.0 (4.24)
  GGT Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  GGT Treatment Course 7, Baseline; n=2 | 14.0 (4.24)
  GGT, Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  GGT, Treatment Course 7, Week 8; n=2 | 14.5 (6.36)
  GGT, Follow-up Week 12; n=59: number analyzed (Participants) | 59
  GGT, Follow-up Week 12; n=59 | 20.5 (18.17)
  GGT, Follow-up Week 24; n=18: number analyzed (Participants) | 18
  GGT, Follow-up Week 24; n=18 | 24.8 (36.99)

26. Secondary Outcome: Assessment of Blood Urea Nitrogen (BUN)
Description: The blood samples of participants were collected to assess the amount of nitrogen (in the form of urea) in the blood. BUN is evaluated to asssess the renal function of the participants.
Time Frame: as for outcome 6
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: millimoles per liter
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
millimoles per liter
  Treatment Course 1, Baseline; n=92 | 5.85 (1.767)
  Treatment Course 1, Week 104; n=1: number analyzed (Participants) | 1
  Treatment Course 1, Week 104; n=1 | 6.40 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Treatment Course 2, Baseline; n=73: number analyzed (Participants) | 73
  Treatment Course 2, Baseline; n=73 | 6.10 (1.781)
  Treatment Course 2, Week 80; n=1: number analyzed (Participants) | 1
  Treatment Course 2, Week 80; n=1 | 9.60 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Treatment Course 3, Baseline; n=53: number analyzed (Participants) | 53
  Treatment Course 3, Baseline; n=53 | 5.78 (1.574)
  Treatment Course 3, Week 64; n=1: number analyzed (Participants) | 1
  Treatment Course 3, Week 64; n=1 | 6.80 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Treatment Course 4, Baseline; n=20: number analyzed (Participants) | 20
  Treatment Course 4, Baseline; n=20 | 5.75 (1.257)
  Treatment Course 4, Week 40; n=1: number analyzed (Participants) | 1
  Treatment Course 4, Week 40; n=1 | 4.60 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  Treatment Course 5, Baseline; n=8: number analyzed (Participants) | 8
  Treatment Course 5, Baseline; n=8 | 5.49 (1.197)
  Treatment Course 5, Week 24; n=2: number analyzed (Participants) | 2
  Treatment Course 5, Week 24; n=2 | 6.05 (0.495)
  Treatment Course 6, Baseline; n=4: number analyzed (Participants) | 4
  Treatment Course 6, Baseline; n=4 | 6.95 (1.700)
  Treatment Course 6, Week 16; n=2: number analyzed (Participants) | 2
  Treatment Course 6, Week 16; n=2 | 7.15 (0.495)
  Treatment Course 7, Baseline; n=2: number analyzed (Participants) | 2
  Treatment Course 7, Baseline; n=2 | 6.60 (0.707)
  Treatment Course 7, Week 8; n=2: number analyzed (Participants) | 2
  Treatment Course 7, Week 8; n=2 | 7.15 (1.061)
  Follow-up Week 12; n=59: number analyzed (Participants) | 59
  Follow-up Week 12; n=59 | 5.79 (1.878)
  Follow-up Week 24; n=18: number analyzed (Participants) | 18
  Follow-up Week 24; n=18 | 6.04 (2.530)

27. Secondary Outcome: Assessment of Systolic Blood Pressure (SBP) and Diastolic Blood Pressure (DBP)
Description: The blood pressure (BP) of the participants was measured before infusion (infu) (BI) and post the first (A) and second (B) infusions (PI) during all 7 treatment courses.Timing for taking BP readings: SBP (BP when the heart is contracting): TC1, 2, 3 (infu A) more than 2 hours PI; TC1, 2 ,3 (infu B) 2 hours PI; TC4, 5, 6, 7 (infu A) 2 hours PI; TC4, 7 (infu B) 2 hours PI; TC5, 6 (infu B) 1 hour PI. For DBP (BP when the heart is resting between beats): TC1, 3 (infu A) more than 2 hours PI; TC2, 4, 5, 6, 7 (infu A) 2 hours PI; TC1, 2, 3, 4, 7 (infu A) 2 hours PI; TC5, 6 (infu B) 1 hour PI.
Time Frame: BI and PI A and B for all TCs (8 wk post infusion, then every 4 wk until Wk 24, then every 8 wk until next treatment course [up to 156 weeks, follow-up phase]). TCs were individualized based on clinical status and may not correlate to trial visits/wk
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: Millimeters of mercury (mmHg)
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
Millimeters of mercury (mmHg)
  SBP, Treatment Course 1, BI-A, n =92 | 121.7 (18.20)
  SBP, Treatment Course 1, PI-A, + >2 Hours, n=2: number analyzed (Participants) | 2
  SBP, Treatment Course 1, PI-A, + >2 Hours, n=2 | 138.5 (3.54)
  SBP, Treatment Course 1, BI-B, n=91: number analyzed (Participants) | 91
  SBP, Treatment Course 1, BI-B, n=91 | 119.9 (18.38)
  SBP, Treatment Course 1, PI-B, + 2 Hours, n=48: number analyzed (Participants) | 48
  SBP, Treatment Course 1, PI-B, + 2 Hours, n=48 | 122.8 (13.22)
  SBP, Treatment Course 2, BI-A, n=73: number analyzed (Participants) | 73
  SBP, Treatment Course 2, BI-A, n=73 | 117.3 (16.84)
  SBP, Treatment Course 2, PI-A, + 2 Hours, n=71: number analyzed (Participants) | 71
  SBP, Treatment Course 2, PI-A, + 2 Hours, n=71 | 121.4 (13.86)
  SBP, Treatment Course 2, BI-B, n=69: number analyzed (Participants) | 69
  SBP, Treatment Course 2, BI-B, n=69 | 116.8 (16.09)
  SBP, Treatment Course 2, PI-B, + 2 Hours, n=36: number analyzed (Participants) | 36
  SBP, Treatment Course 2, PI-B, + 2 Hours, n=36 | 120.5 (13.52)
  SBP, Treatment Course 3, BI-A, n=53: number analyzed (Participants) | 53
  SBP, Treatment Course 3, BI-A, n=53 | 116.8 (15.61)
  SBP, Treatment Course 3, PI-A, + >2 Hours, n=1: number analyzed (Participants) | 1
  SBP, Treatment Course 3, PI-A, + >2 Hours, n=1 | 125.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  SBP, Treatment Course 3, BI-B, n=53: number analyzed (Participants) | 53
  SBP, Treatment Course 3, BI-B, n=53 | 120.1 (15.59)
  SBP, Treatment Course 3, PI-B, + 2 Hours, n=26: number analyzed (Participants) | 26
  SBP, Treatment Course 3, PI-B, + 2 Hours, n=26 | 121.2 (9.63)
  SBP, Treatment Course 4, BI-A, n=20: number analyzed (Participants) | 20
  SBP, Treatment Course 4, BI-A, n=20 | 114.2 (14.86)
  SBP, Treatment Course 4, PI-A, + 2 Hours, n=19: number analyzed (Participants) | 19
  SBP, Treatment Course 4, PI-A, + 2 Hours, n=19 | 116.0 (12.54)
  SBP, Treatment Course 4, BI-B, n=19: number analyzed (Participants) | 19
  SBP, Treatment Course 4, BI-B, n=19 | 111.8 (14.86)
  SBP, Treatment Course 4, PI-B, + 2 Hours, n=2: number analyzed (Participants) | 2
  SBP, Treatment Course 4, PI-B, + 2 Hours, n=2 | 115.0 (15.56)
  SBP, Treatment Course 5, BI-A, n=8: number analyzed (Participants) | 8
  SBP, Treatment Course 5, BI-A, n=8 | 116.1 (16.17)
  SBP, Treatment Course 5, PI-A, + 2 Hours, n=8: number analyzed (Participants) | 8
  SBP, Treatment Course 5, PI-A, + 2 Hours, n=8 | 114.0 (11.99)
  SBP, Treatment Course 5, BI-B, n=8: number analyzed (Participants) | 8
  SBP, Treatment Course 5, BI-B, n=8 | 102.5 (12.54)
  SBP, Treatment Course 5, PI-B, + 1 Hour, n=7: number analyzed (Participants) | 7
  SBP, Treatment Course 5, PI-B, + 1 Hour, n=7 | 103.6 (14.35)
  SBP, Treatment Course 6, BI-A, n=4: number analyzed (Participants) | 4
  SBP, Treatment Course 6, BI-A, n=4 | 123.8 (7.50)
  SBP, Treatment Course 6, PI-A, + 2 Hours, n=4: number analyzed (Participants) | 4
  SBP, Treatment Course 6, PI-A, + 2 Hours, n=4 | 117.5 (12.58)
  SBP, Treatment Course 6, BI-B, n=4: number analyzed (Participants) | 4
  SBP, Treatment Course 6, BI-B, n=4 | 118.8 (13.15)
  SBP, Treatment Course 6, PI-B, + 1 Hour, n=4: number analyzed (Participants) | 4
  SBP, Treatment Course 6, PI-B, + 1 Hour, n=4 | 127.5 (2.89)
  SBP, Treatment Course 7, BI-A, n=2: number analyzed (Participants) | 2
  SBP, Treatment Course 7, BI-A, n=2 | 120.0 (14.14)
  SBP, Treatment Course 7, PI-A, + 2 Hours, n=1: number analyzed (Participants) | 1
  SBP, Treatment Course 7, PI-A, + 2 Hours, n=1 | 125.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  SBP, Treatment Course 7, BI-B, n=2: number analyzed (Participants) | 2
  SBP, Treatment Course 7, BI-B, n=2 | 110.0 (0.00)
  SBP, Treatment Course 7, PI-B, + 2 Hours, n=1: number analyzed (Participants) | 1
  SBP, Treatment Course 7, PI-B, + 2 Hours, n=1 | 125.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  DBP, Treatment Course 1, BI-A, n=92 | 76.3 (11.51)
  DBP, Treatment Course 1, PI-A, +>2 Hours, n=90: number analyzed (Participants) | 90
  DBP, Treatment Course 1, PI-A, +>2 Hours, n=90 | 86.5 (6.36)
  DBP, Treatment Course 1, BI-B, n=91: number analyzed (Participants) | 91
  DBP, Treatment Course 1, BI-B, n=91 | 74.4 (11.85)
  DBP, Treatment Course 1, PI-B, + 2 Hours, n=48: number analyzed (Participants) | 48
  DBP, Treatment Course 1, PI-B, + 2 Hours, n=48 | 75.5 (8.73)
  DBP, Treatment Course 2, BI-A, n=73: number analyzed (Participants) | 73
  DBP, Treatment Course 2, BI-A, n=73 | 73.4 (10.26)
  DBP, Treatment Course 2, PI-A, + 2 Hours, n=71: number analyzed (Participants) | 71
  DBP, Treatment Course 2, PI-A, + 2 Hours, n=71 | 74.8 (8.56)
  DBP, Treatment Course 2, BI-B, n=69: number analyzed (Participants) | 69
  DBP, Treatment Course 2, BI-B, n=69 | 72.8 (10.37)
  DBP, Treatment Course 2, PI-B, + 2 Hours, n=36: number analyzed (Participants) | 36
  DBP, Treatment Course 2, PI-B, + 2 Hours, n=36 | 74.0 (7.58)
  DBP, Treatment Course 3, BI-A, n=53: number analyzed (Participants) | 53
  DBP, Treatment Course 3, BI-A, n=53 | 72.1 (10.84)
  DBP, Treatment Course 3, PI-A, >2 Hours, n=1: number analyzed (Participants) | 1
  DBP, Treatment Course 3, PI-A, >2 Hours, n=1 | 75.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  DBP, Treatment Course 3, BI-B, n=53: number analyzed (Participants) | 53
  DBP, Treatment Course 3, BI-B, n=53 | 74.7 (10.53)
  DBP, Treatment Course 3, PI-B, + 2 Hours, n=26: number analyzed (Participants) | 26
  DBP, Treatment Course 3, PI-B, + 2 Hours, n=26 | 75.3 (8.02)
  DBP, Treatment Course 4, BI-A, n=20: number analyzed (Participants) | 20
  DBP, Treatment Course 4, BI-A, n=20 | 71.7 (11.59)
  DBP, Treatment Course 4, PI-A, + 2 Hours, n=19: number analyzed (Participants) | 19
  DBP, Treatment Course 4, PI-A, + 2 Hours, n=19 | 75.1 (9.79)
  DBP, Treatment Course 4, BI-B, n=19: number analyzed (Participants) | 19
  DBP, Treatment Course 4, BI-B, n=19 | 71.7 (10.87)
  DBP, Treatment Course 4, PI-B, + 2 Hours, n=2: number analyzed (Participants) | 2
  DBP, Treatment Course 4, PI-B, + 2 Hours, n=2 | 75.0 (7.07)
  DBP, Treatment Course 5, BI-A, n=8: number analyzed (Participants) | 8
  DBP, Treatment Course 5, BI-A, n=8 | 74.6 (12.06)
  DBP, Treatment Course 5, PI-A, + 2 Hours, n=8: number analyzed (Participants) | 8
  DBP, Treatment Course 5, PI-A, + 2 Hours, n=8 | 77.5 (10.00)
  DBP, Treatment Course 5, BI-B, n=8: number analyzed (Participants) | 8
  DBP, Treatment Course 5, BI-B, n=8 | 68.4 (6.74)
  DBP, Treatment Course 5, PI-B, +1 Hour, n=7: number analyzed (Participants) | 7
  DBP, Treatment Course 5, PI-B, +1 Hour, n=7 | 69.7 (10.44)
  DBP, Treatment Course 6, BI-A, n=4: number analyzed (Participants) | 4
  DBP, Treatment Course 6, BI-A, n=4 | 77.5 (6.45)
  DBP, Treatment Course 6, PI-A, + 2 Hours, n=4: number analyzed (Participants) | 4
  DBP, Treatment Course 6, PI-A, + 2 Hours, n=4 | 78.8 (4.79)
  DBP, Treatment Course 6, BI-B, n=4: number analyzed (Participants) | 4
  DBP, Treatment Course 6, BI-B, n=4 | 68.8 (10.31)
  DBP, Treatment Course 6, PI-B, 1 Hour, n=4: number analyzed (Participants) | 4
  DBP, Treatment Course 6, PI-B, 1 Hour, n=4 | 81.3 (2.50)
  DBP, Treatment Course 7, BI-A, n=2: number analyzed (Participants) | 2
  DBP, Treatment Course 7, BI-A, n=2 | 85.0 (7.07)
  DBP, Treatment Course 7, PI-A, + 2 Hours, n=1: number analyzed (Participants) | 1
  DBP, Treatment Course 7, PI-A, + 2 Hours, n=1 | 90.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  DBP, Treatment Course 7, BI-B, n=2: number analyzed (Participants) | 2
  DBP, Treatment Course 7, BI-B, n=2 | 75.0 (7.07)
  DBP, Treatment Course 7, PI-B, + 2 Hours, n=1: number analyzed (Participants) | 1
  DBP, Treatment Course 7, PI-B, + 2 Hours, n=1 | 90.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  DBP, Follow-up, n=78: number analyzed (Participants) | 78
  DBP, Follow-up, n=78 | 76.9 (9.16)

28. Secondary Outcome: Assessment of Heart Rate (HR)
Description: The HR of the participants was measured to assess the condition of the heart.HR was measured BI and post the first (A) and second (B) infusins during all 7 treatment courses.Timing for measuring HR: TC1, 3 (infu A) more than 2 hours PI; TC1, 2 ,3, 4, 7 (infu B) 2 hours PI; TC2, 4, 5, 6, 7 (infu A) 2 hours PI; TC5, 6 (infu B) 1 hour PI.
Time Frame: as for outcome 27
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: Beats per minute (bpm)
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
Beats per minute (bpm)
  HR, Treatment Course 1, BI-A, n=92 | 73.4 (10.10)
  HR, Treatment Course 1, PI-A, + >2 Hours, n=2: number analyzed (Participants) | 2
  HR, Treatment Course 1, PI-A, + >2 Hours, n=2 | 76.5 (12.02)
  HR, Treatment Course 1, BI-B, n=91: number analyzed (Participants) | 91
  HR, Treatment Course 1, BI-B, n=91 | 71.8 (9.41)
  HR, Treatment Course 1, PI-B, + 2 Hours, n=48: number analyzed (Participants) | 48
  HR, Treatment Course 1, PI-B, + 2 Hours, n=48 | 74.9 (10.72)
  HR, Treatment Course 2, BI-A, n=73: number analyzed (Participants) | 73
  HR, Treatment Course 2, BI-A, n=73 | 70.9 (7.37)
  HR, Treatment Course 2, PI-A, + 2 Hours, n=71: number analyzed (Participants) | 71
  HR, Treatment Course 2, PI-A, + 2 Hours, n=71 | 74.3 (7.88)
  HR, Treatment Course 2, BI-B, n=69: number analyzed (Participants) | 69
  HR, Treatment Course 2, BI-B, n=69 | 72.9 (8.02)
  HR, Treatment Course 2, PI-B, + 2 Hours, n=36: number analyzed (Participants) | 36
  HR, Treatment Course 2, PI-B, + 2 Hours, n=36 | 73.4 (7.53)
  HR, Treatment Course 3, BI-A, n=53: number analyzed (Participants) | 53
  HR, Treatment Course 3, BI-A, n=53 | 72.6 (6.99)
  HR, Treatment Course 3, PI-A, + >2 Hours, n= 1: number analyzed (Participants) | 1
  HR, Treatment Course 3, PI-A, + >2 Hours, n= 1 | 68.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  HR, Treatment Course 3, BI-B, n=53: number analyzed (Participants) | 53
  HR, Treatment Course 3, BI-B, n=53 | 72.2 (8.57)
  HR, Treatment Course 3, PI-B, + 2 Hours, n=26: number analyzed (Participants) | 26
  HR, Treatment Course 3, PI-B, + 2 Hours, n=26 | 75.6 (6.11)
  HR, Treatment Course 4, BI-A, n=20: number analyzed (Participants) | 20
  HR, Treatment Course 4, BI-A, n=20 | 70.8 (5.77)
  HR, Treatment Course 4, PI-A, + 2 Hours, n=19: number analyzed (Participants) | 19
  HR, Treatment Course 4, PI-A, + 2 Hours, n=19 | 74.6 (6.50)
  HR, Treatment Course 4, BI-B, n=19: number analyzed (Participants) | 19
  HR, Treatment Course 4, BI-B, n=19 | 70.5 (4.43)
  HR, Treatment Course 4, PI-B, + 2 Hours, n=2: number analyzed (Participants) | 2
  HR, Treatment Course 4, PI-B, + 2 Hours, n=2 | 76.0 (5.66)
  HR, Treatment Course 5, BI-A, n=8: number analyzed (Participants) | 8
  HR, Treatment Course 5, BI-A, n=8 | 70.9 (3.00)
  HR, Treatment Course 5, PI-A, + 2 Hours, n=8: number analyzed (Participants) | 8
  HR, Treatment Course 5, PI-A, + 2 Hours, n=8 | 72.6 (3.66)
  HR, Treatment Course 5, BI-B, n=8: number analyzed (Participants) | 8
  HR, Treatment Course 5, BI-B, n=8 | 68.9 (4.58)
  HR, Treatment Course 5, PI-B, + 1 Hour, n=7: number analyzed (Participants) | 7
  HR, Treatment Course 5, PI-B, + 1 Hour, n=7 | 71.7 (4.96)
  HR, Treatment Course 6, BI-A, n=4: number analyzed (Participants) | 4
  HR, Treatment Course 6, BI-A, n=4 | 70.0 (4.00)
  HR, Treatment Course 6, PI-A, + 2 Hours, n=4: number analyzed (Participants) | 4
  HR, Treatment Course 6, PI-A, + 2 Hours, n=4 | 71.0 (6.00)
  HR, Treatment Course 6, BI-B, n=4: number analyzed (Participants) | 4
  HR, Treatment Course 6, BI-B, n=4 | 68.0 (5.66)
  HR, Treatment Course 6, PI-B, + 1 Hour, n=4: number analyzed (Participants) | 4
  HR, Treatment Course 6, PI-B, + 1 Hour, n=4 | 72.0 (0.00)
  HR, Treatment Course 7, BI-A, n=2: number analyzed (Participants) | 2
  HR, Treatment Course 7, BI-A, n=2 | 72.0 (0.00)
  HR, Treatment Course 7, PI-A, + 2 Hours, n=1: number analyzed (Participants) | 1
  HR, Treatment Course 7, PI-A, + 2 Hours, n=1 | 72.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  HR, Treatment Course 7, BI-B, n=2: number analyzed (Participants) | 2
  HR, Treatment Course 7, BI-B, n=2 | 70.0 (2.83)
  HR, Treatment Course 7, PI-B, + 2 Hours, n=1: number analyzed (Participants) | 1
  HR, Treatment Course 7, PI-B, + 2 Hours, n=1 | 68.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  HR, Follow-up, n=78: number analyzed (Participants) | 78
  HR, Follow-up, n=78 | 72.1 (8.05)

29. Secondary Outcome: Assessment of Body Temperature (BT)
Description: The BT of the participants was measured BI and post the first (A) and second (B) infusions (PI) of each cycle to assess the effect of ofatumumab on the BT.The BT of the participants was measured before BI and PI A and B during all 7 treatment courses.Timing for taking BT reading: TC1, 3 (infu A) more than 2 hours PI; TC1, 2 ,3, 4, 7 (infu B) 2 hours PI; TC2, 4, 5, 6, 7 (infu A) 2 hours PI; TC5, 6 (infu B) 1 hour PI.
Time Frame: as for outcome 27
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: Degrees celcius
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
Degrees celcius
  BT, Treatment Course 1, BI-A, n=92 | 36.50 (0.360)
  BT, Treatment Course 1, PI-A, + >2 Hours, n=1: number analyzed (Participants) | 1
  BT, Treatment Course 1, PI-A, + >2 Hours, n=1 | 36.50 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  BT, Treatment Course 1, BI-B, n=91: number analyzed (Participants) | 91
  BT, Treatment Course 1, BI-B, n=91 | 36.46 (0.368)
  BT, Treatment Course 1, PI-B, + 2 Hours, n=48: number analyzed (Participants) | 48
  BT, Treatment Course 1, PI-B, + 2 Hours, n=48 | 36.53 (0.316)
  BT, Treatment Course 2 BI-A, n=73: number analyzed (Participants) | 73
  BT, Treatment Course 2 BI-A, n=73 | 36.48 (0.313)
  BT, Treatment Course 2 PI-A, + 2 Hours, n=71: number analyzed (Participants) | 71
  BT, Treatment Course 2 PI-A, + 2 Hours, n=71 | 36.56 (0.261)
  BT, Treatment Course 2 BI-B, n=69: number analyzed (Participants) | 69
  BT, Treatment Course 2 BI-B, n=69 | 36.54 (0.370)
  BT, Treatment Course 2 PI-B, + 2 Hours, n=36: number analyzed (Participants) | 36
  BT, Treatment Course 2 PI-B, + 2 Hours, n=36 | 36.58 (0.252)
  BT, Treatment Course 3 BI-A, n=53: number analyzed (Participants) | 53
  BT, Treatment Course 3 BI-A, n=53 | 36.46 (0.307)
  BT, Treatment Course 3 PI-A, + >2 Hours, n=1: number analyzed (Participants) | 1
  BT, Treatment Course 3 PI-A, + >2 Hours, n=1 | 36.60 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  BT, Treatment Course 3, BI-B, n=53: number analyzed (Participants) | 53
  BT, Treatment Course 3, BI-B, n=53 | 36.45 (0.392)
  BT, Treatment Course 3, PI-B, + 2 Hours, n=26: number analyzed (Participants) | 26
  BT, Treatment Course 3, PI-B, + 2 Hours, n=26 | 36.59 (0.294)
  BT, Treatment Course 4, BI-A, n=20: number analyzed (Participants) | 20
  BT, Treatment Course 4, BI-A, n=20 | 36.50 (0.381)
  BT, Treatment Course 4, PI-A, + 2 Hours, n=19: number analyzed (Participants) | 19
  BT, Treatment Course 4, PI-A, + 2 Hours, n=19 | 36.58 (0.242)
  BT, Treatment Course 4, BI-B, n=19: number analyzed (Participants) | 19
  BT, Treatment Course 4, BI-B, n=19 | 36.53 (0.421)
  BT, Treatment Course 4, PI-B, + 2 Hours, n=2: number analyzed (Participants) | 2
  BT, Treatment Course 4, PI-B, + 2 Hours, n=2 | 37.00 (0.283)
  BT, Treatment Course 5, BI-A, n=8: number analyzed (Participants) | 8
  BT, Treatment Course 5, BI-A, n=8 | 36.40 (0.267)
  BT, Treatment Course 5, PI-A, + 2 Hours, n=8: number analyzed (Participants) | 8
  BT, Treatment Course 5, PI-A, + 2 Hours, n=8 | 36.50 (0.262)
  BT, Treatment Course 5, BI-B, n=8: number analyzed (Participants) | 8
  BT, Treatment Course 5, BI-B, n=8 | 36.41 (0.242)
  BT, Treatment Course 5, PI-B, + 1 Hour, n=7: number analyzed (Participants) | 7
  BT, Treatment Course 5, PI-B, + 1 Hour, n=7 | 36.49 (0.329)
  BT, Treatment Course 6, BI-A, n=4: number analyzed (Participants) | 4
  BT, Treatment Course 6, BI-A, n=4 | 36.48 (0.126)
  BT, Treatment Course 6, PI-A, + 2 Hours, n=4: number analyzed (Participants) | 4
  BT, Treatment Course 6, PI-A, + 2 Hours, n=4 | 36.48 (0.250)
  BT, Treatment Course 6, BI-B, n=4: number analyzed (Participants) | 4
  BT, Treatment Course 6, BI-B, n=4 | 36.35 (0.370)
  BT, Treatment Course 6, PI-B, + 1 Hour, n=4: number analyzed (Participants) | 4
  BT, Treatment Course 6, PI-B, + 1 Hour, n=4 | 36.45 (0.370)
  BT, Treatment Course 7, BI-A, n=2: number analyzed (Participants) | 2
  BT, Treatment Course 7, BI-A, n=2 | 36.55 (0.071)
  BT, Treatment Course 7, PI-A, + 2 Hours, n=1: number analyzed (Participants) | 1
  BT, Treatment Course 7, PI-A, + 2 Hours, n=1 | 36.60 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  BT, Treatment Course 7, BI-B, n=2: number analyzed (Participants) | 2
  BT, Treatment Course 7, BI-B, n=2 | 36.65 (0.071)
  BT, Treatment Course 7, PI-B, + 2 Hours, n=1: number analyzed (Participants) | 1
  BT, Treatment Course 7, PI-B, + 2 Hours, n=1 | 36.60 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  BT, Follow-up, n=78: number analyzed (Participants) | 78
  BT, Follow-up, n=78 | 36.57 (0.323)

30. Secondary Outcome: Assessment of Lactic Dehydrogenase (LDH) and Creatine Phosphokinase (CPK)
Description: Blood samples of participants were collected to assess LDH and CPK. Both tests are performed to evaluate the injury and damage to the body tissue, potentially from B-cell lysis.
Time Frame: 8 wk post infusion, then every 4 wk until Wk 24, then every 8 wk until next treatment course (up to 144 weeks). TCs were individualized based on clinical status and may not correlate to trial visits or study weeks.
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Mean (Standard Deviation); unit: U/L
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
U/L
  LDH, Treatment Course 1, Baseline, n=92 | 189.6 (35.18)
  LDH, Treatment Course 1, Week 104, n=1: number analyzed (Participants) | 1
  LDH, Treatment Course 1, Week 104, n=1 | 229.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  LDH, Treatment Course 2, Baseline, n=73: number analyzed (Participants) | 73
  LDH, Treatment Course 2, Baseline, n=73 | 198.6 (77.62)
  LDH, Treatment Course 2, Week 80, n=1: number analyzed (Participants) | 1
  LDH, Treatment Course 2, Week 80, n=1 | 219.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  LDH, Treatment Course 3, Baseline, n=53: number analyzed (Participants) | 53
  LDH, Treatment Course 3, Baseline, n=53 | 186.5 (37.39)
  LDH, Treatment Course 3, Week 64, n=1: number analyzed (Participants) | 1
  LDH, Treatment Course 3, Week 64, n=1 | 242.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  LDH, Treatment Course 4, Baseline, n=20: number analyzed (Participants) | 20
  LDH, Treatment Course 4, Baseline, n=20 | 184.6 (35.52)
  LDH, Treatment Course 4, Week 40, n=1: number analyzed (Participants) | 1
  LDH, Treatment Course 4, Week 40, n=1 | 170.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  LDH, Treatment Course 5, Baseline, n=8: number analyzed (Participants) | 8
  LDH, Treatment Course 5, Baseline, n=8 | 179.4 (25.03)
  LDH, Treatment Course 5, Week 24, n=2: number analyzed (Participants) | 2
  LDH, Treatment Course 5, Week 24, n=2 | 168.5 (27.58)
  LDH, Treatment Course 6, Baseline, n=4: number analyzed (Participants) | 4
  LDH, Treatment Course 6, Baseline, n=4 | 173.3 (15.13)
  LDH, Treatment Course 6, Week 16, n=2: number analyzed (Participants) | 2
  LDH, Treatment Course 6, Week 16, n=2 | 234.0 (53.74)
  LDH, Treatment Course 7, Baseline, n=2: number analyzed (Participants) | 2
  LDH, Treatment Course 7, Baseline, n=2 | 292.0 (140.01)
  LDH, Treatment Course 7, Week 8, n=2: number analyzed (Participants) | 2
  LDH, Treatment Course 7, Week 8, n=2 | 190.0 (25.46)
  CPK, Treatment Course 1, Baseline, n=92 | 61.4 (29.25)
  CPK, Treatment Course 1, Week 104, n=1: number analyzed (Participants) | 1
  CPK, Treatment Course 1, Week 104, n=1 | 127.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CPK, Treatment Course 2, Baseline, n=73: number analyzed (Participants) | 73
  CPK, Treatment Course 2, Baseline, n=73 | 70.5 (31.07)
  CPK, Treatment Course 2, Week 80, n=1: number analyzed (Participants) | 1
  CPK, Treatment Course 2, Week 80, n=1 | 61.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CPK, Treatment Course 3, Baseline, n=53: number analyzed (Participants) | 53
  CPK, Treatment Course 3, Baseline, n=53 | 77.7 (50.86)
  CPK, Treatment Course 3, Week 64, n=1: number analyzed (Participants) | 1
  CPK, Treatment Course 3, Week 64, n=1 | 81.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CPK, Treatment Course 4, Baseline n=20: number analyzed (Participants) | 20
  CPK, Treatment Course 4, Baseline n=20 | 85.4 (64.46)
  CPK, Treatment Course 4, Week 40, n=1: number analyzed (Participants) | 1
  CPK, Treatment Course 4, Week 40, n=1 | 52.0 (NA) — Standard deviation is not calculated when only one participant was analyzed.
  CPK, Treatment Course 5, Baseline, n=8: number analyzed (Participants) | 8
  CPK, Treatment Course 5, Baseline, n=8 | 157.6 (216.71)
  CPK, Treatment Course 5, Week 24, n=2: number analyzed (Participants) | 2
  CPK, Treatment Course 5, Week 24, n=2 | 82.5 (27.58)
  CPK, Treatment Course 6, Baseline, n=4: number analyzed (Participants) | 4
  CPK, Treatment Course 6, Baseline, n=4 | 84.8 (23.91)
  CPK, Treatment Course 6, Week 16, n=2: number analyzed (Participants) | 2
  CPK, Treatment Course 6, Week 16, n=2 | 100.0 (14.14)
  CPK, Treatment Course 7, Baseline, n=2: number analyzed (Participants) | 2
  CPK, Treatment Course 7, Baseline, n=2 | 103.0 (19.80)
  CPK, Treatment Course 7, Week 8, n=2: number analyzed (Participants) | 2
  CPK, Treatment Course 7, Week 8, n=2 | 109.0 (15.56)
  CPK, Follow-up Week 12, n=59: number analyzed (Participants) | 59
  CPK, Follow-up Week 12, n=59 | 79.3 (38.73)
  CPK, Follow-up Week 24, n=18: number analyzed (Participants) | 18
  CPK, Follow-up Week 24, n=18 | 77.0 (26.09)

31. Secondary Outcome: Number of Participants With Normal and Abnormal Electrocardiogram Readings
Description: Electrocardiograms of the participants were taken. The abnormal clinically significant (CS) and not clinically significant (NCS) reading, as determined by the Investigator, were recorded.
Time Frame: as for outcome 30
Population: FAS Population. Only participants with data available at particular time points were analyzed.
Measure: Number; unit: participants
Arm/Group | Ofatumumab 700 mg IV Infusion
Number analyzed (Participants) | 92
participants
  Treatment Course 1, Week 24, Normal | 64
  Treatment Course 1, Week 24, Abnormal NCS | 9
  Treatment Course 1, Week 24, Abnormal CS | 0
  Treatment Course 1, Week 104, Normal | 1
  Treatment Course 1, Week 104, Abnormal NCS | 0
  Treatment Course 1, Week 104, Abnormal CS | 0
  Treatment Course 2, Week 24, Normal | 43
  Treatment Course 2, Week 24, Abnormal NCS | 17
  Treatment Course 2, Week 24, Abnormal CS | 0
  Treatment Course 2, Week 80, Normal | 1
  Treatment Course 2, Week 80, Abnormal NCS | 0
  Treatment Course 2, Week 80, Abnormal CS | 0
  Treatment Course 3, Week 24, Normal | 24
  Treatment Course 3, Week 24, Abnormal NCS | 4
  Treatment Course 3, Week 56, Normal | 1
  Treatment Course 3, Week 56, Abnormal NCS | 1
  Treatment Course 3, Week 56, Abnormal CS | 0
  Treatment Course 4, Week 24, Normal | 7
  Treatment Course 4, Week 24, Abnormal NCS | 0
  Treatment Course 4, Week 24, Abnormal CS | 0
  Treatment Course 4, Week 32, Normal | 3
  Treatment Course 4, Week 32, Abnormal NCS | 0
  Treatment Course 4, Week 32, Abnormal CS | 0
  Treatment Course 5, Week 24, Normal | 2
  Treatment Course 5, Week 24, Abnormal NCS | 0
  Treatment Course 5, Week 24, Abnormal CS | 0

ADVERSE EVENTS:
Arm/Group | Ofatumumab 700 mg IV Infusion
Serious Adverse Events (participants affected / at risk) | 11/92
Other Adverse Events (participants affected / at risk) | 70/92
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab 700 mg IV Infusion (N=92)
Memory impairment (Nervous system disorders) | 2
Amnesia (Nervous system disorders) | 1
Aphasia (Nervous system disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Disturbance in attention (Nervous system disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Hypertension (Vascular disorders) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Myocardial infarction (Cardiac disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Pneumonia (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 1
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 1
Visual impairment (Eye disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab 700 mg IV Infusion (N=92)
Upper respiratory tract infection (Infections and infestations) | 14
Rhinitis (Infections and infestations) | 5
Urinary tract infection (Infections and infestations) | 5
Bronchitis (Infections and infestations) | 4
Nasopharyngitis (Infections and infestations) | 4
Oral herpes (Infections and infestations) | 4
Influenza (Infections and infestations) | 3
Pharyngitis (Infections and infestations) | 3
Respiratory tract infection (Infections and infestations) | 3
Sinusitis (Infections and infestations) | 3
Abscess (Infections and infestations) | 2
Cystitis (Infections and infestations) | 2
Lower respiratory tract infection (Infections and infestations) | 2
Enterobiasis (Infections and infestations) | 1
Eye infection (Infections and infestations) | 1
Furuncle (Infections and infestations) | 1
Gastroenteritis viral (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Lobar pneumonia (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Rash pustular (Infections and infestations) | 1
Skin infection (Infections and infestations) | 1
Tonsillitis (Infections and infestations) | 1
Tracheitis (Infections and infestations) | 1
Rash (Skin and subcutaneous tissue disorders) | 20
Urticaria (Skin and subcutaneous tissue disorders) | 5
Pruritus (Skin and subcutaneous tissue disorders) | 3
Alopecia (Skin and subcutaneous tissue disorders) | 2
Rash generalized (Skin and subcutaneous tissue disorders) | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1
Erythema (Skin and subcutaneous tissue disorders) | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 1
Rash erythematous (Skin and subcutaneous tissue disorders) | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 10
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 9
Sneezing (Respiratory, thoracic and mediastinal disorders) | 6
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 5
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 3
Dry throat (Respiratory, thoracic and mediastinal disorders) | 2
Throat tightness (Respiratory, thoracic and mediastinal disorders) | 2
Bronchospasm (Respiratory, thoracic and mediastinal disorders) | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 1
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1
Nasal dryness (Respiratory, thoracic and mediastinal disorders) | 1
Pharyngeal edema (Respiratory, thoracic and mediastinal disorders) | 1
Postnasal drip (Respiratory, thoracic and mediastinal disorders) | 1
Rhinorrhea (Respiratory, thoracic and mediastinal disorders) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2
Bursitis (Musculoskeletal and connective tissue disorders) | 2
Rheumatoid arthritis (Musculoskeletal and connective tissue disorders) | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 1
Flank pain (Musculoskeletal and connective tissue disorders) | 1
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1
Limb discomfort (Musculoskeletal and connective tissue disorders) | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Sensation of heaviness (Musculoskeletal and connective tissue disorders) | 1
Spondylolisthesis (Musculoskeletal and connective tissue disorders) | 1
Synovial cyst (Musculoskeletal and connective tissue disorders) | 1
Tendon disorder (Musculoskeletal and connective tissue disorders) | 1
Headache (Nervous system disorders) | 9
Aphasia (Nervous system disorders) | 3
Memory impairment (Nervous system disorders) | 3
Disturbance in attention (Nervous system disorders) | 2
Hypoaesthesia (Nervous system disorders) | 2
Sciatica (Nervous system disorders) | 2
Amnesia (Nervous system disorders) | 1
Dysgeusia (Nervous system disorders) | 1
Meralgia paraesthetica (Nervous system disorders) | 1
Neuralgia (Nervous system disorders) | 1
Paraesthesia (Nervous system disorders) | 1
Nausea (Gastrointestinal disorders) | 3
Diarrhea (Gastrointestinal disorders) | 2
Dry mouth (Gastrointestinal disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Periodontitis (Gastrointestinal disorders) | 2
Abdominal distension (Gastrointestinal disorders) | 1
Dental caries (Gastrointestinal disorders) | 1
Duodenal ulcer (Gastrointestinal disorders) | 1
Mouth ulceration (Gastrointestinal disorders) | 1
Pancreatitis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 1
Hepatic enzyme Increased (Investigations) | 3
Alanine aminotransferase increased (Investigations) | 2
Aspartate aminotransferase increased (Investigations) | 2
Blood creatinine increased (Investigations) | 2
Blood alkaline phosphatase increased (Investigations) | 1
Blood immunoglobulin G decreased (Investigations) | 1
Blood pressure increased (Investigations) | 1
Blood urea increased (Investigations) | 1
Blood uric acid increased (Investigations) | 1
Cardiac murmur (Investigations) | 1
Heart rate abnormal (Investigations) | 1
John Cunningham virus test positive (Investigations) | 1
Neutrophil count decreased (Investigations) | 1
Transaminases increased (Investigations) | 1
Neutropenia (Blood and lymphatic system disorders) | 5
Leukopenia (Blood and lymphatic system disorders) | 4
Anemia (Blood and lymphatic system disorders) | 3
Lymphopenia (Blood and lymphatic system disorders) | 2
Lymphadenopathy (Blood and lymphatic system disorders) | 1
Conjunctivitis (Eye disorders) | 3
Dry eye (Eye disorders) | 3
Visual impairment (Eye disorders) | 2
Conjunctival irritation (Eye disorders) | 1
Eye swelling (Eye disorders) | 1
Eyelid edema (Eye disorders) | 1
Lacrimation increased (Eye disorders) | 1
Photopsia (Eye disorders) | 1
Vision blurred (Eye disorders) | 1
Visual acuity reduced (Eye disorders) | 1
Vitreous floaters (Eye disorders) | 1
Hypertension (Vascular disorders) | 4
Flushing (Vascular disorders) | 3
Varicophlebitis (Vascular disorders) | 1
Varicose vein (Vascular disorders) | 1
Fall (Injury, poisoning and procedural complications) | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1
Limb crushing injury (Injury, poisoning and procedural complications) | 1
Patella fracture (Injury, poisoning and procedural complications) | 1
Tendon rupture (Injury, poisoning and procedural complications) | 1
Upper limb fracture (Injury, poisoning and procedural complications) | 1
Fatigue (General disorders) | 4
Edema peripheral (General disorders) | 2
Chest discomfort (General disorders) | 1
Influenza like illness (General disorders) | 1
Thirst (General disorders) | 1
Vertigo (Ear and labyrinth disorders) | 3
Ear pruritus (Ear and labyrinth disorders) | 1
Tinnitus (Ear and labyrinth disorders) | 1
Atrial fibrillation (Cardiac disorders) | 1
Myocardial infarction (Cardiac disorders) | 1
Tachycardia (Cardiac disorders) | 1
Oral allergy syndrome (Immune system disorders) | 2
Allergy to vaccine (Immune system disorders) | 1
Fluid retention (Metabolism and nutrition disorders) | 1
Gout (Metabolism and nutrition disorders) | 1
Hyperuricemia (Metabolism and nutrition disorders) | 1
Increased appetite (Metabolism and nutrition disorders) | 1
Anxiety (Psychiatric disorders) | 1
Depression (Psychiatric disorders) | 1
Insomnia (Psychiatric disorders) | 1
Stress (Psychiatric disorders) | 1
Leukocyturia (Renal and urinary disorders) | 1
Nephrolithiasis (Renal and urinary disorders) | 1
Nocturia (Renal and urinary disorders) | 1
Proteinuria (Renal and urinary disorders) | 1
Renal impairment (Renal and urinary disorders) | 1
Demoid cyst (Congenital, familial and genetic disorders) | 1
Cholecystitis (Hepatobiliary disorders) | 1
Cholelithiasis (Hepatobiliary disorders) | 1
Seborrhoeic keratosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1
Breast pain (Reproductive system and breast disorders) | 1

LIMITATIONS AND CAVEATS:
Development of the IV route of ofatumumab (OFA) administration in RA will no longer be pursued. This study was prematurely terminated; OFA treatment was discontinued. Participants could complete only <=7 treatment courses and a follow-up evaluation.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.